Division: World Wide Development Retention Category: GRS019

Information Type: Reporting and Analysis Plan

Title: Reporting and Analysis Plan for AMB114588:

> An open-label, long term extension study for treatment of pulmonary arterial hypertension in paediatric patients aged 8 years up to 18 years who have participated in AMB112529 and

in whom continued treatment with ambrisentan is desired.

Compound Number: GSK1325760

Effective Date: 03 Jun 2022

**Description**: This document outlines the safety and efficacy reporting planned for

protocol AMB114588 by GlaxoSmithKline (GSK).

Identifier/Version Number: Version 2.0

Subject: GSK1325760, Pulmonary Arterial Hypertension, Long Term Extension,

Paediatrics; Reporting, Tables, Figures, Listings (TFLs)

PPD Author's Name, Title and Functional Area: PPD

Hartington Statistics and Data Management Ltd.

Updates by PPD

Approved by:

Senior Manager-Statistics Development Statistics

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| AB | BREVI | ATIONS . | | 5 |
| 1. | INTR | ODUCTIO | DN | 7 |
| _ | OTLIE | ) | OTIVE(O) AND ENDROINT(O) | - |
| 2. | 2.1. | Other C | CTIVE(S) AND ENDPOINT(S) | / |
| | 2.1. | 2.1.1. | Objective(s)Primary Objective | |
| | | 2.1.1. | Secondary Objectives | |
| | 2.2. | | indpoint(s) | |
| | | 2.2.1. | · | |
| | | 2.2.2. | | |
| | | | 2.2.2.1. Pharmacokinetics | 8 |
| | | | 2.2.2.2. Efficacy | 8 |
| | | | 2.2.2.3. Exploratory | |
| | | a | 2.2.2.4. Other | |
| | 2.3. | | cal Hypotheses | |
| | 2.4. | Pnarma | cokinetic (PK) and PK/Pharmacodynamic (PD) hypotheses | 9 |
| 3. | STUE | Y DESIG | N | 9 |
| 4. | PLAN | INED ANA | ALYSES | 9 |
| | 4.1. | | Analyses | |
| | 4.2. | Final Ar | nalysis | 9 |
| 5. | SAMF | PLE SIZE | CONSIDERATIONS | 9 |
| 6. | ANAL | YSIS PO | PULATIONS | 10 |
| 7. | TREA | TMENT ( | COMPARISONS | 10 |
| | 7.1. | | splay Treatment and Other Sub-group Descriptors | |
| 8. | GENE | ERAL CO | NSIDERATIONS FOR DATA ANALYSES | 10 |
| | 8.1. | | ation of Subgroups | |
| 9. | DATA | HANDLI | NG CONVENTIONS | 10 |
| | 9.1. | Premati | ure Withdrawal and Missing Data | |
| | | 9.1.1. | Missing Efficacy Outcomes Data | |
| | | 9.1.2. | Missing AE data | 11 |
| | | 9.1.3. | Missing Dates (other than for AEs) | |
| | 0.2 | 9.1.4. | Missing Items on SF-10 | |
| | 9.2. | 9.2.1. | and Transformed DataBaseline | |
| | | 9.2.1. | Change from baseline and percentage change from | 12 |
| | | J.Z.Z. | baselinebaseline and percentage change from | 12 |
| | | 9.2.3. | WHO FC change from baseline categorisation 1 | |
| | | 9.2.4. | WHO FC class change from baseline categorisation 2 | |
| | | 9.2.5. | Study Day | 13 |
| | | 9.2.6. | Age Calculation | 13 |

| | | 9.2.7. Duration of Exposure | 13 |
|---|---|---|---|
| | | 9.2.8. Transformations for Efficacy Outcomes | 13 |
| | | 9.2.9. Treatment Compliance Rates | |
| | 9.3. | Assessment Windows | |
| | 9.4. | Values of Clinical Concern | |
| | | 9.4.1. Laboratory Parameters | |
| | | 9.4.2. Vital Signs | |
| 10. | STUD | Y POPULATION | 16 |
| | 10.1. | Disposition of Subjects | |
| | 10.2. | Protocol Deviations | |
| | 10.3. | Medical Conditions | 17 |
| | 10.4. | Prior and Concomitant Medications | 17 |
| | 10.5. | Treatment Compliance | 17 |
| 11. | SAFE | TY ANALYSES | 18 |
| | 11.1. | Extent of Exposure | 18 |
| | 11.2. | | |
| | 11.3. | Adverse Events Leading to Discontinuation of Investigational | |
| | | Product and/or Withdrawal from the Study and Other Significant | |
| | | Adverse Events | |
| | 11.4. | Deaths and Serious Adverse Events | |
| | 11.5. | Adverse Events of Special Interest | |
| | 11.6. | Non-serious Adverse Events | |
| | 11.7. | Laboratory Evaluations | |
| | | 11.7.1. Liver Events | |
| | | 11.7.2. Vital Signs | |
| | 44.0 | 11.7.3. Physical Examination | |
| | 11.8. | 12-Lead ECG. | |
| | 11.9. | | |
| | | Change in dose due to tolerability issues | |
| | 11.11. | Pregnancies (as applicable) | 21 |
| <b>12</b> . | | ACY ANALYSES | |
| | 12.1. | | |
| | 12.2. | Other analyses | 22 |
| 13. | | TIONAL ANALYSES DUE TO THE COVID-19 PANDEMIC | |
| | 13.1 | Study Population | |
| | | 13.2 Subject Disposition and Protocol Deviations | |
| | | 13.3 Protocol Deviations | 23 |
| | | 13.4 Additional Displays for Participants with a COVID-19 Infection | 22 |
| | | 13.5 Additional Analyses Due to the COVID-19 Pandemic | 23<br>29 |
| | | 13.6 Assessment of COVID-19 AEs | |
| 14. | | CAL PHARMACOLOGY DATA ANALYSES | |
| | 14.1. | Pharmacokinetic Analyses | |
| | 14.2. | | |
| | 14.3. | Pharmacokinetic/Pharmacodynamic Analyses | 24 |
| 15 | BIOM | ARKER DATA ANALYSIS | 24 |

| 16. | PHARMACOGENETIC DATA ANALYSES | 24 |
|-----|-------------------------------|----------------|
| 17. | VIRAL GENOTYPING/PHENOTYPING | 24 |
| 18. | REFERENCES | 24 |
| 19. | ATTACHMENTS | 25<br>31<br>34 |
| 20. | APPENDICES | |

# **ABBREVIATIONS**

| 6MWD | 6 minute walking distance test |
|------------|----------------------------------------------|
| AE | Adverse Event |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body mass index |
| BSA | Body surface area |
| DBF | Database Freeze |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| FC | Functional Class |
| GGT | gamma glutamyl transferase |
| GSK | GlaxoSmithKline |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| ITT | Intent-to-Treat |
| kg | Kilogram |
| m | Meter |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| NT-Pro BNP | N-Terminal pro-B-type Natriuretic Peptide |
| PAH | Pulmonary Arterial Hypertension |
| PD | Pharmacodynamic |
| PDE-5 | Phosphodiesterase type 5 |
| PHS | Physical Summary |
| PK | Pharmacokinetic |
| PSS | Psychosocial Summary |
| PT | Preferred Term |
| RA | Right atrial |
| RV | Right ventricle |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Ststem |
| SD | Standard Deviation |
| SF | Short Form |
| SOC | System Organ Class |
| TAPSE | Tricuspid annular plane systolic excursion |
| TEAE | Treatment-emergent adverse events |
| TRJ | Tricuspid regurgitant jet |
| ULN | Upper limit of normal |
| WHO | World Health Organization |

5

# **Trademark Information**

| Trademarks of the GlaxoSmithKline group of companies |
|------------------------------------------------------|
| AMBRISENTAN |
| FLOLAN |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| Adcirca |
| C RIBA |
| Letairis |
| NONMEM |
| Remodulin |
| Revatio |
| Thelin |
| Tracleer |
| Ventavis |
| Viagra |

#### 1. INTRODUCTION

This Reporting and Analysis Plan (RAP) outlines the safety and efficacy reporting planned for protocol AMB114588 for provision to GSK.

In this RAP, reference is made to the protocol AMB114588 dated 8<sup>th</sup> February 2011, and subsequent amendments.

# 2. STUDY OBJECTIVE(S) AND ENDPOINT(S)

# 2.1. Study Objective(s)

This final RAP was updated following Protocol Amendment 4, in which the study was brought to early closure prior to the remaining active subjects either completing 18 years of treatment (1 subject) and/or having a pubertal assessment at 20 years of age.

# 2.1.1. Primary Objective

The primary objective of this study is to evaluate the long term safety and tolerability of ambrisentan in the paediatric (aged 8 years up to 18 years) PAH population.

# 2.1.2. Secondary Objectives

The secondary objective is to obtain supportive efficacy data (change from baseline in efficacy parameters) on the paediatric use of ambrisentan in PAH.

# 2.2. Study Endpoint(s)

# 2.2.1. Primary Endpoints

- Adverse Events;
- Serious Adverse Events;
- Clinical laboratory parameters;
- Physical examination (including height, weight, body mass index / body surface area, oxygen saturation, jugular venous pressure, liver size, and presence of peripheral oedema and/or ascites);
- Vital Signs;
- Pubertal development (change from Study AMB112529 baseline in endocrinology assessments every six months and at 20 years of age unless pubertal maturity has been reached in previous visits)
- The time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to tolerability issues (e.g. adverse events).

## 2.2.2. Secondary Endpoints

#### 2.2.2.1. Pharmacokinetics

Not applicable.

# 2.2.2.2. Efficacy

- All cause mortality;
- The change from Study AMB112529 baseline in the 6 minute walking distance (6MWD) test evaluated every six months;
- The time to clinical worsening of PAH;
- The time to addition of another targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to the following reasons:
  - Deterioration of clinical condition;
  - Lack of beneficial effect with previous therapy (not reaching set treatment goals);
- The time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition;
- The change from Study AMB112529 baseline in Subject Global Assessment every three months using the SF-10 health survey for children;
- The change from Study AMB112529 baseline in WHO functional class every six months;
- Change from Study AMB112529 baseline in N-terminal pro-B-type natriuretic peptide (NT-Pro BNP) concentration every six months.
- School days missed due to PAH.

#### 2.2.2.3. Exploratory

• The change from Study AMB112529 baseline in major prognostic factors based on echocardiogram: pericardial effusion, right atrial (RA) pressure, tricuspid annular plane systolic excursion (TAPSE), eccentricity index (systolic and diastolic), and right ventricular (RV) pressure by tricuspid regurgitant jet (TRJ) velocity at every 6 months.

#### 2.2.2.4. Other

• The change from Study AMB112529 baseline in cardiopulmonary hemodynamic assessments data in subjects in whom hemodynamic data is considered part of the standard of care.

# 2.3. Statistical Hypotheses

No formal hypothesis is planned.

# 2.4. Pharmacokinetic (PK) and PK/Pharmacodynamic (PD) hypotheses

Not applicable.

#### 3. STUDY DESIGN

This is an open label, long term extension to Study AMB112529. All subjects may remain in the extension study for a minimum of six months. Beyond the six month period, subjects may continue in the extension study until one of the following conditions is met:

- The subject turns 18 years of age (when the subject can receive marketed product). or the subject has reached pubertal maturity before 18 years of age and ambrisentan can be supplied through a named patient or expanded access program until the subject reaches 18 years of age;
- The product is approved and available for use in the subject's age group;
- Development for use in the paediatric population is discontinued;
- The subject decides he/she no longer wants to participate in the study;
- The investigator considers it is in the best interest of the subject to discontinue ambrisentan (e.g. for safety reasons).

Protocol waivers or exemptions are not allowed. Therefore, adherence to the study design requirements, including those specified in the Time and Events Table, are essential. For further details regarding the study design, please refer to the protocol.

#### 4. PLANNED ANALYSES

# 4.1. Interim Analyses

An interim analysis was added post the finalization of the study protocol, in order to provide analyses in support of regulatory interactions. All data collected by a predetermined clinical cut-off date will be analyzed as per this RAP for the interim analysis report.

# 4.2. Final Analysis

This analysis plan outlines the final analysis that will be performed on the safety and efficacy endpoints of this study, once Database Freeze (DBF) has taken place.

# 5. SAMPLE SIZE CONSIDERATIONS

Sample size is based on feasibility. Due to low prevalence of the disease, no more than 66 subjects will be enrolled in the study. No sample size sensitivity calculations were performed. No sample size re-estimation is planned.

#### 6. ANALYSIS POPULATIONS

The Intention-to-Treat (ITT) Population will consist of all subjects who received at least 1 dose of study drug. For the ITT population, subjects were considered as belonging to their treatment group at the start of study AMB114588. The ITT population will be used in all efficacy summaries.

The Safety Population is defined as all subjects who received at least 1 dose of study drug. Subjects were considered as belonging to the treatment group according to the highest dose received. The Safety Population will be used in all safety summaries.

The Idiopathic Group Population is defined as subjects having an Idiopathic Aetiology of PAH (IPAH) at start of study treatment in AMB112529.

## 7. TREATMENT COMPARISONS

There are no formal comparisons planned for this study. Doses of ambrisentan will be summarized descriptively based on available data.

# 7.1. Data Display Treatment and Other Sub-group Descriptors

Refer to the data display specification in Section 19 for examples showing how treatment groups will be displayed in the study report data displays.

## 8. GENERAL CONSIDERATIONS FOR DATA ANALYSES

All programming of tables, figures and listings will be performed using Statistical Analysis System (SAS®) version 8.2 or higher.

# 8.1. Examination of Subgroups

Selected safety and efficacy outputs will be produced by age strata (8-11, 12-18 years).

Selected outputs will also be produced for patients enrolled at centres in Japan to support registration activities.

#### 9. DATA HANDLING CONVENTIONS

All data displays will be presented according to the GSK's Integrated Data Standards Library (IDSL) statistical display principles. The file extension used for landscape tables and listings will be L10, with point size of 10, line size of 108 and 43 lines per page. Where data are sparse, empty tables may be produced with the "Data too sparse for table to be produced" or "No Data to Report" or similar.

All data collected on the electronic case report form (eCRF) will be listed. Data collected outside of the eCRFs (eg. labs, SF10) will also be listed. All listings will be presented by treatment group and subject identification number.

# 9.1. Premature Withdrawal and Missing Data

Subjects who withdraw from the study will not be replaced and all information obtained from them will be included in the summaries.

# 9.1.1. Missing Efficacy Outcomes Data

No imputation will be made for any missing numerical data, unless otherwise specified.

Missing data will generally not be considered in the calculation of percentages (i.e., the denominator will not include subjects who have missing data at a given time point).

## 9.1.2. Missing AE data

Where a start date for an adverse event (AE) is partial or missing, the following imputation rules will be applied:

- If day portion is missing, set day to 1.
- If month portion is missing, set month to January.
- If the date is completely missing, or if the date imputed using the above rules is prior to the first dose date, set the date to first dose date.

Where an end date for an AE is partial or missing, the following imputation rules will be applied. These will only be applied to AEs that are resolved; if they are not resolved then nothing will be imputed.

- If day portion is missing, set day to the last day of the month.
- If month portion is missing, set month to December.
- If the date is completely missing, or if the date imputed using the above rules is after the treatment end date, set the date to the treatment end date or if the treatment end date is missing then set to date of discontinuation.

No further imputation will be performed for missing data.

# 9.1.3. Missing Dates (other than for AEs)

For any data type that collects partial dates, impute missing day as 01 and missing month as January. If date is completely missing then date should remain missing. Where the start date of study medication is missing, the date of randomisation will be used. Where end date of study medication is partial or missing, the last complete non-missing date of dosing will be used as the last date for determining duration of exposure.

#### 9.1.4. Missing Items on SF-10

The SF-10 will be scored in accordance with the developer's guidelines. Out-of-range values are converted to missing values and no algorithm is used to estimate missing values. The Physical and Psychosocial summary scores are not calculated if any component scores are missing.

#### 9.2. Derived and Transformed Data

All listings will include all subjects that have the relevant data for each listing. The number of subjects (N) in each treatment group and overall for the population being summarised, will be displayed in each table unless specified otherwise. For continuous data, the following summary statistics will be presented: n, mean, standard deviation (SD), median, upper and lower quartiles, minimum and maximum. Mean and median values will be reported to one decimal place greater than the original data they were collected from while the SD will be reported to two decimal places greater than the original data however, if this results in a value of 0.00 being presented then a zero (0) will be presented. Minimum and maximum values will be reported with the same precision as they were collected.

All text fields must be left justified. Numeric or numeric with some text specification (e.g., not done, unknown, <4.5, ...) must be right justified.

The format for dates will be DDMMMYYYY.

All tables and listings will have the protocol number and population in the top left-hand corner and the page number in the form of page x of n will be presented in the top right-hand corner. In the bottom left-hand corner of tables and listings the name of the person who created the output followed by a colon, the output filepath and the date and time of the production of the output, in the form DDMMMYYYY HH:MM, will be displayed. If a count in a table summary is zero (0) then a percentage will not be presented. To determine whether an adverse event is on-treatment and a medication is prior or concomitant, imputation of missing or partial start and stop dates is required (see RAP Section 9.1.2 and Section 9.1.3). Imputed dates will not be listed and adverse event duration will not be calculated if the start date or stop date had to be imputed.

#### 9.2.1. Baseline

Baseline values are those collected prior to the first dose (from Study AMB112529). Therefore, if a subject has no data for a parameter on Day 1 (prior to first dose) then the data from their last pre-treatment assessment will be used.

# 9.2.2. Change from baseline and percentage change from baseline

For untransformed data change from baseline at Week X will be calculated as Week X value minus baseline value. The percentage change from baseline at Week X will be calculated as:  $100 \times (\text{Week X value} - \text{baseline value}) / \text{baseline value}$ .

For log-transformed data (see Section 9.2.8), ratio to baseline expressed as percentage change will be calculated by taking the mean change on the log scale, exponentiating, subtracting 1 and multiplying by 100.

(Exp(mean of (Log x - Log baseline)) -1)\*100

## 9.2.3. WHO FC change from baseline categorisation 1

Note that based on the study inclusion criteria subjects must have a WHO FC of II or III at baseline. Change from baseline at Week X will be calculated as Week X value minus baseline value, thus categories may be -2, -1, 0, +1, +2.



## 9.2.4. WHO FC class change from baseline categorisation 2

in Change from Baseline Categorisation
in Change from Baseline Categorisation
in Change from Baseline Categorisation

# 9.2.5. Study Day

Study Day 1 is defined as the day of the first dose of study drug in AMB112529.

Relative Day to start of study medication for an Event is defined as:

Date of event - Date of first study medication + 1, if the event is on or after the first dose date.

Date of event - Date of first study medication, if the event is prior to the first dose date. Relative Day to end of medication for an Event is defined as:

Date of event - Date of last study medication + 1, if the event is on or after the last dose date.

Date of event - Date of last study medication, if the event is prior to the last dose date.

#### 9.2.6. Age Calculation

Age in years at baseline will be derived as a whole number according to the IDSL standard algorithm (see Appendix 1).

#### 9.2.7. Duration of Exposure

Duration of exposure will be calculated in days as (Treatment stop date – Treatment start date in AMB112529) + 1.

#### 9.2.8. Transformations for Efficacy Outcomes

A log transformation will be applied to NT-proBNP data.

Summaries of the relative changes from baseline based on analysis of log-transformed data will include the geometric mean and coefficient of variation (calculated as below based on the logged values) and the geometric mean of the ratio of the value of the endpoint at the time point of interest to the baseline value (see Section 9.2.2).

Geometric mean =  $\exp(\mu)$ 

Coefficient of variation =s  $100 \times \sqrt{\exp(\sigma^2) - 1}$ 

## 9.2.9. Treatment Compliance Rates

Compliance to study medication is recorded at each visit in one of the following categorical groups:

- 0% compliant (subject did not take any doses)
- >0% and < 80% compliant (subject missed a number of doses)
- >=80% and <=120%, (number of doses taken was within compliance range)
- >120% compliant (number of doses taken exceeds compliance limits)

At the subject level compliance rate is calculated as 100\* (the number of visits at which the subject was compliant (i.e.  $\geq 80\%$  and  $\leq 120\%$ ) / (the sum of all study visits for the subject).

At a treatment group level compliance rate is calculated as 100\* (the total number of visits at which all subjects in that group were compliant (i.e.  $\geq$  80% and  $\leq$  120%)) / (the sum of all study visits for all subjects in that group).

#### 9.3. Assessment Windows

All data will be reported for the whole study period.

Unscheduled assessments will not be slotted to a particular time point, but will remain as unscheduled unless otherwise specified.

Time points relating to nominal visits will be used in tables, figures and listings.

Time to clinical worsening of PAH and time to liver event will be calculated using the date of assessment.

#### 9.4. Values of Clinical Concern

# 9.4.1. Laboratory Parameters

The following values of potential clinical concern will be considered:

| Values of potential clinical concern values will be defined for laboratory parameters as follows: Parameter | Code | Units | Low<br>Concern<br>Value (SI<br>units) | High<br>Concern<br>Value (SI<br>units) | Worse case direction |
|---|---|---|---|---|---|
| Hematology | | | | | |
| Hemoglobin | HGB | G/L | Males: < 98 Females: < 91 | Males: > 180.0<br>Females: > 161.0 | Low |

| Values of potential clinical concern values will be defined for laboratory parameters as follows: Parameter | Code | Units | Low<br>Concern<br>Value (SI<br>units) | High<br>Concern<br>Value (SI<br>units) | Worse case direction |
|---|---|---|---|---|---|
| Hematocrit | НСТ | %<br>(1) | Males:<br>< 32.0<br>(<0.32)<br>Females:<br><29.0<br>(<0.29) | Males: > 54.0 (>0.54) Females: > 50.6 (>0.506) | Low |
| Platelets | PLATE | 10^9/L<br>(same as<br>GI/L) | < 100 | > 500 | Low |
| Chemistry | | | | | |
| Total bilirubin | BILTOT | UMOL/L | None | >= 34.2 | High |
| AST | ASAT | IU/L | None | >= 3 x<br>ULN | High |
| ALT | ALAT | IU/L | None | >= 3 x<br>ULN | High |
| GGT | GGT | IU/L | None | >= 3 x<br>ULN | High |
| Creatinine | CREAT | UMOL/L | None | >= 176.8 | High |

## 9.4.2. Vital Signs

The following criteria will be used to determine whether a subject's vital signs (blood pressure and heart rate) lie outside a pre-determined range of clinical concern:

| Parameter | Code | Units | Low Concern<br>Value | High Concern Value |
|---|---|---|---|---|
| Heart Rate | PUL | Bpm | < 50 | > 120 |
| Systolic | SYS | mm Hg | < 80 | > 160 mm Hg<br>> 30 mm Hg change from<br>Baseline |
| Diastolic | DIA | mm Hg | < 40 | > 110 mm Hg<br>> 20 mm Hg change from<br>Baseline |
| Body weight | WT | Kg | < 20 | |

# 10. STUDY POPULATION

Study population data will be presented for the Intent-to-Treat Population unless otherwise specified.

# 10.1. Disposition of Subjects

The number of subjects eligible for each of the analysis populations will be summarised by treatment group and overall, and by country and centre.

The number of subjects completing/withdrawing from the study along with the reasons for withdrawal will be summarised by treatment group and overall.

#### 10.2. Protocol Deviations

The number of subjects with important protocol deviations will be summarised by treatment group and overall.

A summary of subjects who did not satisfy all inclusion and exclusion criteria will be provided by treatment group.

The protocol deviations will be reviewed by the clinical team after the database release and prior to the database freeze, to determine which ones are considered to be important Demographic and Baseline Characteristics.

The number and percentage of subjects in each category for categorical variables or summary statistics for continuous variables will be summarised by treatment group and overall. These include age, age strata, sex, child-bearing potential, ethnicity and geographic ancestry, aetiology of PAH strata, duration of PAH, PAH therapy use, WHO FC score and 6 minute walk distance.

#### 10.3. Medical Conditions

The number and percentage of subjects with past or current medical conditions will be summarised by treatment group and overall, for any condition and by condition classification.

#### 10.4. Prior and Concomitant Medications

The GSKdrug dictionary will be used to code drug names.

Prior medications are those that started and stopped prior to the date of first study treatment. Ongoing medications at baseline are those started before first dose date of study drug, which were continued during the treatment phase.

Lab medications are defined as:

- Medications that start prior to or on the date of first study treatment and that stopped prior to the date of last study treatment,
- Medications that start prior to or on the date of first study treatment and continued after the date of last study treatment,
- Medications that start after the date of first study treatment and that stopped prior to the date of the last study treatment,
- Medications that start after the date of first study treatment and continued after the date of last study treatment.

Any medications that started after the last study treatment are classed as post-treatment medications.

Note that it will be assumed that the medication has been taken by the medication start and stop dates recorded in the eCRF.

The number and percentage of subjects with concomitant medications will be summarised by Anatomical Therapeutic Chemical (ATC) Classification System code and drug name Preferred term by treatment group and overall.

The number and percentage of subjects with ongoing (at entry to AMB114588) and concomitant PAH therapy (at 6 months after entry into AMB114588 and then annually as well as the final visit) will be summarised by preferred term, by treatment group and overall. The ATC codes from the GSKDrug dictionary for the groupings of PAH therapy will be agreed with the Clinical Safety Group and provided in a separate file. This includes:

- PDE5i
- Prostanoid

# 10.5. Treatment Compliance

Every three months, treatment compliance will be recorded as 0%, >0% - <80%, =>80% - <=120% and >120%.

The number and percentage of subjects in each compliance category will be summarised at each visit by treatment group and overall.

# 11. SAFETY ANALYSES

Safety data will be presented for the Safety Population unless otherwise specified.

# 11.1. Extent of Exposure

The number of days of exposure to study drug will be summarised by treatment group and overall.

This number of days of exposure will be categorised in 30 day intervals as follows: <=30 days, 31-60 days, 61-90 days etc.

The number and percentage of subjects in each of these categories will be summarised by treatment group and overall.

#### 11.2. Adverse Events

All AEs will be categorised into Preferred Term (PT) and associated System Organ Class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary.

Only treatment-emergent adverse events (TEAEs) will be included in summary tables. TEAEs are defined as those events that start on or after first dose date of study treatment. Any subject with at least one reported TEAE will be classified as a subject with:

- A TEAE,
- A TEAE leading to study treatment discontinuation (definitive or temporary),
- A TEAE leading to study withdrawal,
- At least one serious TEAE.

The numbers and percentages of subjects with at least one reported TEAE will be summarised by treatment group and overall according to:

- PT,
- SOC and PT,
- SOC and PT by intensity,
- SOC and PT by relationship to study treatment,
- PT by action taken with investigational product (IP).

Recurring TEAEs (i.e. successive TEAEs classified with the same PT) for a given subject will only be counted once and only their most severe intensity will be tabulated. The cumulative incidence of each TEAE will also be summarised by SOC and PT and the following categories: <=3 months, >3 to <=6months, etc.

TEAEs will be listed by SOC and PT, by treatment with the number of subjects who experienced the event and their subject numbers presented. A more detailed listing will also be produced for all subjects who experienced an AE.

# 11.3. Adverse Events Leading to Discontinuation of Investigational Product and/or Withdrawal from the Study and Other Significant Adverse Events

The numbers and percentages of subjects with at least one reported TEAE leading to discontinuation of the investigational product or withdrawal from the study will be summarised by SOC and PT for each treatment group and overall. Covid-19 adverse event data will be shown here if any exist.

#### 11.4. Deaths and Serious Adverse Events

Summary tables detailed in sections 11.2 and Section 11.3 (with the exception of cumulative incidence) will be repeated for serious TEAEs.

Summary tables will also be presented for serious TEAEs by PT and outcome for each treatment group and overall.

A summary of serious TEAEs displaying the number of subjects and occurrences will also be presented.

In addition, the number of subjects with fatal TEAEs and fatal TEAEs related to IP will be summarised by SOC and PT for each treatment group and overall.

# 11.5. Adverse Events of Special Interest

Summary tables detailed in sections 11.2 and Section 11.3 (with the exception of tables by maximum intensity/grade, action taken and relation to IP) will be repeated for AEs of special interest. MedDRA preferred terms and codes for AEs of special interest will be agreed with Clinical Safety Group and provided in a separate file.

The adverse events of special interest are:

- Anaemia
- Hepatoxicity
- Hypersensitivity
- Hypotension
- Male infertility
- Oedema
- Fluid retention

#### 11.6. Non-serious Adverse Events

A summary of the most common (>=5%) non-serious TEAEs displaying the number of subjects and occurrences will also be presented.

# 11.7. Laboratory Evaluations

Absolute values and changes from baseline of laboratory data will be summarised for each visit, by treatment group and overall.

Separate tables will be presented for haematology data, clinical chemistry data and endocrine data (females only).

The number and percentages of subjects with laboratory values above and below reference ranges for potential clinical concern described in Section 9.4.1 will be summarised for each visit, by treatment group and overall.

#### 11.7.1. Liver Events

The number and percentage of subjects reporting a liver event will be summarised: overall, during and post study treatment.

The following will be listed by treatment group, for subjects with liver events:

- liver chemistry result involved in the event.
- Time from first and last dose to start of event
- Patient specific information for liver events
- Medical conditions.
- Liver biopsy details.
- Liver imaging details.

# 11.7.2. Vital Signs

Absolute values and changes from baseline of vital signs data will be summarised for each visit, by treatment group and overall.

The number and percentages of subjects with vital signs values or change from baseline values above and below reference ranges for potential clinical concern described in Section 9.4.2 will be summarised for each visit, by treatment group and overall.

#### 11.7.3. Physical Examination

Physical examination at each visit will be summarised by treatment group and overall.

#### 11.8. 12-Lead ECG

The number and percentages of subjects with electrocardiogram (ECG) abnormalities (clinically significant and not clinically significant) will be summarised for each visit, by treatment group and overall.

# 11.9. Endocrinology

The following will be summarised for each visit (as appropriate) by treatment group and overall.

- Female breast development and pubic hair development.
- Male testicular volume, genital development and pubic hair development.
- Change from baseline in male testicular volume.
- Change from baseline in plasma endocrine parameters (Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B) by gender.

The above tables will also be summarised by pubertal status at baseline defined as follows:

Male: Pre-pubertal: testicular volume < 4 ml, Post-pubertal: testicular volume  $\ge 4$  ml. Female: Pre-pubertal: Stage 1 breast development, Post-pubertal: Stage  $\ge 2$  breast development.

# 11.10. Change in dose due to tolerability issues

The time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to tolerability issues (e.g. adverse events) will be summarised by treatment group and overall.

# 11.11. Pregnancies (as applicable)

A listing of pregnancy events will be provided, as necessary.

# 12. EFFICACY ANALYSES

Efficacy data will be presented for the Intent-to-Treat Population unless otherwise specified.

The following will be summarised for observed case data for each visit (as appropriate) by treatment group and overall.

- All cause mortality.
- The absolute value, change from Study AMB112529 baseline and % change from baseline in the 6 minute walking distance (6MWD) test, overall and by oxygen use.
- The walking duration for subjects who walked less than six minutes.
- The use of oxygen during the 6MWD test.
- The time to clinical worsening of PAH.
- The criteria for clinical worsening of PAH.
- The time to addition of another targeted PAH therapeutic agent (prostanoids, PDE-5 inhibitors) due to the following reasons:
  - o Deterioration of clinical condition;
  - Lack of beneficial effect with previous therapy (not reaching set treatment goals);
- The time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition.
- WHO Functional Class and change from Study AMB112529 baseline in WHO Functional Class.
- The absolute value and percent change from Study AMB112529 baseline, using log-transformed data, in N-terminal pro-B-type natriuretic peptide (NT-Pro BNP) concentration.
- The absolute value and change from baseline in the number of school days, missed school days and missed school days due to PAH.
- The absolute value and change from Study AMB112529 baseline in Subject Global Assessment as measured by the SF-10 health survey for children and summarised for the physical summary score (PHS-10) and the psychosocial summary score (PSS-10).

Further table will be produced summarizing change in WHO FC scores categorized in terms of and in terms of Section 9.2.3 and Section 9.2.4).

# 12.1. Exploratory analyses

The following will be summarised for each visit, by treatment group and overall.

 The absolute value and change from Study AMB112529 baseline in exploratory echocardiogram: pericardial effusion, right atrial pressure, tricuspid annular plane systolic excursion, eccentricity index (systolic and diastolic), tricuspid regurgitant jet velocity and right ventricular pressure.

# 12.2. Other analyses

The following will be listed for each visit, by treatment group.

The absolute value and change from Study AMB112529 baseline in cardiopulmonary hemodynamics (at centres where the collection of hemodynamic data is considered part of the standard of care):- heart rate, mean arterial blood pressure, mean pulmonary arterial pressure, mean right atrial pressure, left ventricular end diastolic pressure or pulmonary capillary wedge pressure, pulmonary vascular resistance, cardiac output, cardiac index (calculated value), arterial oxygen saturation and mixed venous oxygen saturation.

# 13. ADDITIONAL ANALYSES DUE TO THE COVID-19 PANDEMIC

# 13.1 Study Population

No changes required as enrollment was completed at time of COVID-19 restrictions.

# 13.2 Subject Disposition and Protocol Deviations

A country level listing of the dates of the COVID-19 Pandemic measures will be produced, as well as a listing of visits impacted by the COVID-19 Pandemic.

#### Phases of COVID-19 Pandemic Measures

Pandemic measures began in different countries at different times. A dataset containing the date when pandemic measures began, as determined by the GSK country Issue Management Teams (IMT), will be used to determine the start date of pandemic measures within each country. A copy of this dataset will be taken at the time of database freeze (DBF).

The 'Summary of Subject Status and Subject Disposition for the Study Conclusion Record' and the 'Summary of Treatment Status and Reasons for Discontinuation of Study Treatment' will be repeated, with the reason for withdrawal/discontinuation categorised as due to the COVID-19 pandemic, or non-due to the COVID-19 pandemic based on information collected on the COVID-19 Pandemic Study Impact form.

#### 13.3 Protocol Deviations

In addition to the overall summary of important protocol deviations, a separate summary will be produced of important protocol deviations related to COVID-19.

# 13.4 Additional Displays for Participants with a COVID-19 Infection

A participant is defined as having a suspected, probable or confirmed COVID-19 infection during the study if the answer is "Confirmed", "Probable" or "Suspected" to the case diagnosis question from the COVID-19 coronavirus infection assessment eCRF. Summaries and/or listings of the numbers of participants with a suspected, probable or confirmed COVID-19 infection, and of COVID-19 test results will be presented.

# 13.5 Additional Analyses Due to the COVID-19 Pandemic

Visits and assessments missed due to the COVID-19 pandemic, together with visits conducted remotely, will be summarised in a table and listed by subject. The summaries will be based on GSK Core Data Standards, and details are provided in Section 4: List of Data Displays.

#### 13.6 Assessment of COVID-19 AEs

A terms of interest list, list code 319259, created by the GSK dictionaries group, will be used to identify all COVID-19 AEs.

The incidence of AEs and SAEs (Fatal and Non-Fatal) of COVID-19, COVID-19 AEs leading to study drug discontinuation, and COVID-19 AEs leading to study withdrawal, and COVID-19 AEs by severity, will be obtained from standard AE and SAE summaries if data exist to meet the criteria. A listing of relevant data will be created.

# 14. CLINICAL PHARMACOLOGY DATA ANALYSES

# 14.1. Pharmacokinetic Analyses

Not applicable.

# 14.2. Pharmacodynamic Analyses

Not applicable.

# 14.3. Pharmacokinetic/Pharmacodynamic Analyses

Not applicable.

#### 15. BIOMARKER DATA ANALYSIS

Not applicable.

#### 16. PHARMACOGENETIC DATA ANALYSES

Not applicable.

#### 17. VIRAL GENOTYPING/PHENOTYPING

Not applicable.

#### 18. REFERENCES

# 19. ATTACHMENTS

# 19.1. Table of Contents for Data Display Specifications

# 19.1.1. Tables

Table numbering for the Japanese subgroup will be add 001 at the end of the table number. Thus, Table 1.1 will become 1.1001. Table numbering for the Age Strata subgroup will be add 002 at the end of the table number. Thus, Table 1.5 will become 1.5002.

Japanese and Age subgroup analysis will not be needed for final SAC.

Population Tables

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age strata subgroup analysis | Deliverable |
|---|---|---|---|---|---|---|
| 1.1 | Summary of Subject Disposition (See 2 additional rows added to existing table: 1) additional row 20 year count, and 1 covid death related row) Prog Note: The deaths should be mutually exclusive (ie only in 1 category) | Intent-to-<br>Treat | 1.1 | X | unarysis | Interim, SAC |
| 1.2 | Summary of Study Populations | Randomised | 1.2 | | | Interim, SAC |
| 1.3 | Summary of Subjects by Country and Centre | Intent-to-<br>Treat | 1.3 | | Disclosure | Interim, SAC |
| 1.4 | Summary of Inclusion/Exclusion Criteria Deviations | Intent-to-<br>Treat | 1.4 | | | Interim, SAC |
| 1.5 | Summary of Demographic and Baseline Characteristics | Intent-to-<br>Treat | 1.5 | Х | X | Interim, SAC |
| 1.6 | Summary of Past Medical Conditions | Intent-to-<br>Treat | 1.6 | | X | Interim, SAC |
| 1.7 | Summary of Current Medical Conditions | Intent-to-<br>Treat | 1.6 | | X | Interim, SAC |
| 1.8 | Summary of Concomitant Medications | Intent-to-<br>Treat | 1.8 | Х | | Interim, SAC |
| 1.9 | Summary of Ongoing Background PAH Therapy at Entry Visit to AMB114588 By Drug Class and Preferred Term | Intent-to-<br>Treat | 1.9 | | X | Interim, SAC |
| 1.10 | Summary of Ongoing Background PAH Therapy by Drug<br>Class and Preferred Term | Intent-to-<br>Treat | 1.9 | | X | Interim, SAC |
| 1.11 | Summary of Compliance to Investigational Product since last visit | Intent-to-<br>Treat | 1.11 | | | Interim, SAC |
| 1.12 | Summary of Investigational Product Compliance Overall | Intent-to-<br>Treat | 1.12 | | | Interim, SAC |
| 1.13 | Summary of initial dose of ambrisentan at entry to AMB114588 and highest dose received during study | Intent-to-<br>Treat | 1.13 | | | Interim, SAC |
| 1.14 | Summary of initial dose of ambrisentan at entry to AMB114588 and final dose at end of study or termination | Intent-to-<br>Treat | 1.14 | | | Interim, SAC |
| 1.15 | Summary of Important Protocol Deviation | Intent-to-<br>Treat | 1.15 | | | Interim, SAC |
| 1.16 | Summary of Concomitant Medications starting in AMB114588 | Intent-to-<br>treat | 1.8 | | | Added at<br>Interim |

|--|

| Table<br>Number | Title | Population | Template<br>Table | Deliverable | Programming Notes |
|---|---|---|---|---|---|
| 1.17 | Summary of Important<br>COVID-19 Related<br>Protocol Deviations | Intent-to-<br>Treat | Same as protocol DV table except subset for COVID-19 related | SAC [1] | |
| 1.18 | Summary of COVID-19 Assessments for Subjects with Suspected, Probable or Confirmed COVID-19 Case Diagnosis | Intent-to-<br>Treat | 1.19 | SAC [1] | |
| 1.19 | Summary of Visits impacted by COVID-19 Pandemic | Intent-to-<br>Treat | 1.20 | SAC [1] | |

Efficacy Tables

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 2.1 | Summary of Time to Death (All cause) (days) | Intent-to-<br>Treat | 2.1 | X | X | Interim, SAC |
| 2.2 | Summary of 6 Minute Walking Distance (meters) | Intent-to-<br>Treat | 2.2 | Х | X | Interim, SAC |
| 2.3 | Summary of Change from Baseline in 6 Minute Walking Distance (meters) | Intent-to-<br>Treat | 2.2 | X | X | Interim, SAC |
| 2.4 | Summary of Percent Change from Baseline in 6 Minute Walking Distance (meters) | Intent-to-<br>Treat | 2.2 | Х | X | Interim, SAC |
| 2.5 | Summary of Walking Duration (minutes) for subjects who walked less than six minutes | Intent-to-<br>Treat | 2.5 | X | X | Interim, SAC |
| 2.6 | Summary of use of Oxygen during 6 Minute Walking exercise (L/min) | Intent-to-<br>Treat | 2.6 | X | X | Interim, SAC |
| 2.7 | Summary of Time to Clinical Worsening of PAH (days) | Intent-to-<br>Treat | 2.7 | X | | Interim, SAC |
| 2.8 | Summary of Clinical Worsening of PAH | Intent-to-<br>Treat | 2.8 | | | Interim, SAC |
| 2.9 | Summary of Time to the addition of another targeted PAH therapeutic agent (prostanoids, PDE-5 inhibitors) (days) | Intent-to-<br>Treat | 2.9 | X | | Interim, SAC |
| 2.10 | Summary of Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition (days) | Intent-to-<br>Treat | 2.10 | Х | | Interim, SAC |
| 2.11 | Summary of WHO Functional Class | Intent-to-<br>Treat | 2.11 | Х | X | Interim, SAC |
| 2.12 | Summary of Change from Baseline in WHO Functional Class | Intent-to-<br>Treat | 2.11 | Х | X | Interim, SAC |
| 2.13 | Summary of WHO Functional Class Shifts from Baseline by Visit | Intent-to-<br>Treat | 2.13 | Х | X | Interim, SAC |
| 2.14 | Summary of WHO Functional Class Change from Baseline Categorisation | Intent-to-<br>Treat | 2.14 | X | X | Interim, SAC |
| 2.15 | Summary of Plasma NT-Pro BNP concentration (ng/L) | Intent-to-<br>Treat | 2.15 | X | X | Interim, SAC |
| 2.16 | Summary of Ratio to Baseline in Plasma NT-Pro BNP concentration (%) | Intent-to-<br>Treat | 2.15 | Х | X | Interim, SAC |

|-----|--------------|-----------|

| Table | Title | Population | Template | Japanese | Age | Deliverable |
|---|---|---|---|---|---|---|
| Number | | | Table | subgroup<br>analysis | strata<br>subgroup<br>analysis | |
| 2.17 | Summary of Exploratory Echocardiogram | Intent-to-<br>Treat | 2.17 | Х | X | Interim, SAC |
| 2.18 | Summary of Change from Baseline in Exploratory Echocardiogram | Intent-to-<br>Treat | 2.18 | X | X | Interim, SAC |
| 2.19 | Summary of Number of Subjects with School Days | Intent-to-<br>Treat | 2.19 | Х | X | Interim, SAC |
| 2.20 | Summary Statistics of School Days | Intent-to-<br>Treat | 2.20 | Х | X | Interim, SAC |
| 2.21 | Summary Statistics of Change from Baseline in School Days | Intent-to-<br>Treat | 2.20 | Х | X | Interim, SAC |
| 2.22 | Summary of Subject Global Assessment (SF10 Health Survey for Children) | Intent-to-<br>Treat | 2.22 | Х | X | Interim, SAC |
| 2,23 | Summary of Change from Baseline in Subject Global Assessment (SF10 Health Survey for Children) | Intent-to-<br>Treat | 2.22 | Х | X | Interim, SAC |
| 2.24 | Summary of SF10 Health Survey - Number and Percentage of Subjects with Particular Item Responses | Intent-to-<br>Treat | 2.24 | X | X | Interim, SAC |
| 2.25 | Number of subjects who achieved a clinically significant improvement (20 Meters) in 6 min walk | Intent-to-<br>Treat | 2.25 | | | GSK SAC,<br>Internal |
| 2.26 | Number of subjects who achieved a clinically significant improvement (20 Meters) in 6 min walk | Idiopathic<br>Group | 2.26 | | | GSK SAC,<br>Internal |
| 2.27 | Number of subjects who achieved an NT-proBNP levels of less than 1200 ng/L | Intent-to-<br>Treat | 2.27 | | | GSK SAC,<br>Internal |
| 2.28 | Number of subjects who achieved an NT-proBNP levels of less than 1200 ng/L | Idiopathic<br>Group | 2.28 | | | GSK SAC,<br>Internal |
| 2.29 | Distribution of NT-proBNP levels at baseline and extent of change during treatment | Intent-to-<br>Treat | 2.29 | | | GSK SAC,<br>Internal |
| 2.30 | Distribution of NT-proBNP levels at baseline and extent of change during treatment | Idiopathic<br>Group | 2.30 | | | GSK SAC,<br>Internal |
| 2.31 | The Event Rate of the Clinical Worsening Endpoint per 100 Patient-Years | Intent-to-<br>Treat | 2.31 | | | GSK SAC,<br>Internal |

# Safety Tables

| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age strata subgroup analysis | Deliverable |
|---|---|---|---|---|---|---|
| 3.1 | Summary of Exposure to Investigational Product <b>New Footnote:</b> For subjects missing their last exposure date at the time of study end, their last visit date in the study was used. | Safety | 3.1 | Х | Х | Interim, SAC |
| 3.2 | Summary of Treatment-Emergent Adverse Events | Safety | 3.2 | X | X | Interim, SAC |
| 3.3 | Summary of Treatment-Emergent Adverse Events by Preferred Term | Safety | 3.3 | | X | Interim, SAC |
| 3.4 | Summary of Treatment-Emergent Adverse Events by Maximum Intensity | Safety | 3.4 | Х | | Interim, SAC |
| 3.5 | Summary of Treatment-Emergent Adverse Events by Action Taken with IP | Safety | 3.5 | | | Interim, SAC |

| RAP | | / | CONFIDENTIAL | | | | AMB11458 |
|---|---|---|---|---|---|---|---|
| Table | Title | | Population | Template | e Japanese | Age strata | Deliverable |
| Number | | | | Table | subgroup | subgroup | |
| | | | | | analysis | analysis | |

| Table | Title | Population | Template | Japanese | Age strata | Deliverable |
|---|---|---|---|---|---|---|
| Number | | | Table | subgroup<br>analysis | subgroup<br>analysis | |
| 3.6 | Summary of Treatment-Emergent Adverse Events leading to Permanent Discontinuation of IP or Withdrawal from the Study | Safety | 3.2 | | Х | Interim, SAC |
| 3.7 | Summary of Treatment-Emergent Adverse Events related to IP | Safety | 3.2 | Х | X | Interim, SAC |
| 3.8 | Summary of Cumulative Incidence of Treatment-<br>Emergent Adverse Events by Time to First Occurrence | Safety | 3.8 | | | Interim, SAC |
| 3.9 | Summary of Serious Treatment-Emergent Adverse<br>Events | Safety | 3.2 | | X | Interim, SAC |
| 3.10 | Summary of Serious Treatment-Emergent Adverse<br>Events - Number of Subjects and Occurrences | Safety | 3.10 | | Disclosure | Interim, SAC |
| 3.11 | Summary of Serious Treatment-Emergent Adverse<br>Events by Outcome | Safety | 3.11 | | | Interim, SAC |
| 3.12 | Summary of Serious Treatment-Emergent Adverse<br>Events by Action Taken with IP | Safety | 3.5 | | | Interim, SAC |
| 3.13 | Summary of Serious Treatment-Emergent Adverse<br>Events leading to Permanent Discontinuation of IP<br>or Withdrawal from the Study | Safety | 3.2 | | | Interim, SAC |
| 3.14 | Summary of Serious Treatment-Emergent Adverse<br>Events related to IP | Safety | 3.2 | | Disclosure | Interim, SAC |
| 3.15 | Summary of Fatal Serious Treatment-Emergent Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.16 | Summary of Fatal Serious Treatment-Emergent Adverse Events related to IP | Safety | 3.2 | | Disclosure | Interim, SAC |
| 3.17 | Summary of Treatment-Emergent Adverse Events of Special Interest | Safety | 3.2 | X | | Interim, SAC |
| 3.18 | Summary of Treatment-Emergent Adverse Events of<br>Special Interest leading to Permanent<br>Discontinuation of IP or Withdrawal from the Study | Safety | 3.2 | | | Interim, SAC |
| 3.19 | Summary of Cumulative Incidence of Treatment-<br>Emergent Adverse Events of Special Interest by Time<br>to First Occurrence | Safety | 3.8 | | | Interim, SAC |
| 3.20 | Summary of Most Common (>5%) Non-Serious Treatment-<br>Emergent Adverse Events - Number of Subjects and<br>Occurrences | Safety | 3.10 | | Disclosure | Interim, SAC |
| 3.21 | Summary of Haematology Data | Safety | 3.21 | X | | Interim, SAC |
| 3.22 | Summary of Change from Baseline in Haematology Data | Safety | 3.21 | X | | Interim, SAC |
| 3.23 | Summary of Haematology Data of Potential Clinical Concern | Safety | 3.23 | X | | Interim, SAC |
| 3.24 | Summary of Clinical Chemistry Data | Safety | 3.21 | X | | Interim, SAC |
| 3.25 | Summary of Change from Baseline in Clinical<br>Chemistry Data | Safety | 3.21 | X | | Interim, SAC |
| 3.26 | Summary of Clinical Chemistry Data of Potential Clinical Concern | Safety | 3.23 | X | | Interim, SAC |
| 3.27 | Summary of Endocrinology Laboratory Data (females only) | Safety | 3.21 | X | | Interim, SAC |
| 3.28 | Summary of Change from Baseline in Endocrinology Laboratory Data (females only) | Safety | 3.21 | X | | Interim, SAC |
| 3.29 | Summary of Liver Events Assessment | Safety | 3.29 | | | Interim, SAC |

| RAP | / cc | NFIDENTIAL | | | | AMB11458 |
|---|---|---|---|---|---|---|
| | | | 1 | | | |
| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age strata subgroup analysis | Deliverable |
| 3.30 | Summary of Vital Signs | Safety | 3.30 | X | | Interim, SAC |
| 3.31 | Summary of Change from Baseline in Vital Signs | Safety | 3.30 | X | | Interim, SAC |
| 3.32 | Summary of Vital Signs Data of Potential Clinical Concern | Safety | 3.32 | X | | Interim, SAC |
| 3.33 | Summary of Change from Baseline in Vital Signs Da-<br>of Potential Clinical Concern | ta Safety | 3.32 | X | | Interim, SAC |
| 3.34 | Summary of Physical Examination by Visit | Safety | 3.34 | Х | | Interim, SAC |
| 3.35 | Summary of 12-lead ECG | Safety | 3.35 | Х | | Interim, SAC |
| 3.36 | Summary of Endocrinology assessments by Visit - Female | Safety | 3.36 | х | ADDED: Footnote re 20 year assessments in all TLF's | Interim, SAC |
| 3.37 | Summary of Endocrinology assessments by Visit - Male | Safety | 3.37 | Х | ADDED: Footnote | Interim, SAC |
| 3.38 | Summary of Pubertal Development Shifts from Baseline - Female | Safety | 3.38 | X | ADDED:<br>Footnote | Interim, SAC |
| 3.39 | Summary of Pubertal Development Shifts from Baseline - Male | Safety | 3.39 | X | ADDED:<br>Footnote | Interim, SAC |
| 3.40 | Summary of Testicular Volume Change from Baseline Male | - Safety | 3.40 | X | ADDED:<br>Footnote | Interim, SAC |
| 3.41 | Summary of Change from Baseline in Plasma Endocrip<br>Parameters - Female | ne Safety | 3.41 | Х | ADDED:<br>Footnote | Interim, SAC |
| 3.42 | Summary of Change from Baseline in Plasma Endocrin<br>Parameters - Male | ne Safety | 3.42 | Х | ADDED:<br>Footnote | Interim, SAC |
| 3.43 | Summary of Time to change in dose of ambrisentan other targeted PAH therapeutic agents (prostanoid PDE-5 inhibitors) due to tolerability issues (day | s, | 2.10 | X | | Interim, SAC |
| 3.44 | Summary of Treatment Emergent Adverse Events Starting in AMB114588 | | 3.44 | | | SAC |
| 3.45 | Summary of Treatment Emergent Adverse Events by PAH Therapy | Safety | 3.44 | | | GSK SAC,<br>Internal S&P |
| 3.46 | Summary of Serious Treatment Emergent Adverse<br>Events by PAH Therapy | e Safety | 3.44 | | | GSK SAC,<br>Internal S&P |
| 3.47 | Summary of Non-Serious Treatment Emergent Adverse Events by PAH Therapy | Safety | 3.44 | | | GSK SAC,<br>Internal S&P |
| 3.48 | Summary of Common (>=5%) Treatment Emergent Adverse Events by PAH Therapy | Safety | 3.44 | | | GSK SAC,<br>Internal S&P |
| | Footnote: Note: Common adverse events (>=5%) were those experienced by at least 5% of subjects in the total population (N=38) irrespective of dose group and/or PAH therapy | | | | | |
| 3.49 | Summary of Treatment Emergent Adverse Events by PAH Aetiology | Safety | 3.48 | | | GSK SAC,<br>Internal S&P |

| RAP | CONE | FIDENTIAL | | | | AMB114588 |
|---|---|---|---|---|---|---|
| Table<br>Number | Title | Population | Template<br>Table | Japanese<br>subgroup<br>analysis | Age strata<br>subgroup<br>analysis | Deliverable |
| 3.50 | Summary of Serious Treatment Emergent Adverse<br>Events by PAH Aetiology | Safety | 3.48 | | | GSK SAC,<br>Internal S&P |
| 3.51 | Summary of non-Serious Treatment Emergent Adverse Events by PAH Aetiology | Safety | 3.48 | | | GSK SAC,<br>Internal S&P |
| 3.52 | Summary of Common (>=5%) Treatment Emergent Adverse Events by PAH Aetiology Footnote: Note: Common adverse events (>=5%) were those experienced by at least 5% of subjects in the total population (N=38) irrespective of dose group and/or PAH Aetiology. | Safety | 3.48 | | | GSK SAC,<br>Internal S&P |
| 3,53 | Summary of Cardiopulmonary Hemodynamics | Safety | 3.52 | | | SAC-New |

# 19.1.2. **Listings**

# Population Listings

| Listing<br>Number | Title | Population | Template<br>Listing | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 1.1 | Listing of Reasons for Study Withdrawal | Intent-to-<br>Treat | 1.1 | | | Interim, SAC |
| 1.2 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | Intent-to-<br>Treat | 1.2 | | | Interim, SAC |
| 1.3 | Listing of Demographic Characteristics | Intent-to-<br>Treat | 1.3 | | | Interim, SAC |
| 1.4 | Listing of Race | Intent-to-<br>Treat | 1.4 | | | Interim, SAC |
| 1/.5 | Listing of Disease History | Intent-to-<br>Treat | 1.5 | | | Interim, SAC |
| 1.6 | Listing of Medical Conditions | Intent-to-<br>Treat | 1.6 | | | Interim, SAC |
| 1.7 | Listing of Medications | Intent-to-<br>Treat | 1.7 | | | Interim, SAC |
| 1.8 | Listing of PAH Therapy | Intent-to-<br>Treat | 1.8 | | | Interim, SAC |
| 1.9 | Relationship between ATC Level 1, Ingredient and Verbatim Text | Intent-to-<br>Treat | 1.9 | | | Interim, SAC |
| 1.10 | Listing of Compliance Data | Intent-to-<br>Treat | 1.10 | | | Interim, SAC |
| 1.11 | Listing of initial, highest and final dose of ambrisentan | Intent-to-<br>Treat | 1.11 | | | |
| 1.12 | Listing of Protocol Deviation | Intent-to-<br>Treat | 1.12 | | | Interim, SAC |

Efficacy Listings

| Listing | Title | Population | Template | Japanese | Age | Deliverable |
|---|---|---|---|---|---|---|
| Number | | | Listing | subgroup<br>analysis | strata<br>subgroup<br>analysis | |
| 2.1 | Listing of Time to Death (All cause) | Intent-to-<br>Treat | 2.1 | | | Interim, SAC |
| 2.2 | Listing of 6 Minute Walking Distance Data | Intent-to-<br>Treat | 2.2 | | | Interim, SAC |
| 2.3 | Listing of Clinical Worsening of PAH | Intent-to-<br>Treat | 2.3 | | | Interim, SAC |
| 2.4 | Listing of Time to the addition of another targeted PAH therapeutic agent (prostanoids, PDE-5 inhibitors) | Intent-to-<br>Treat | 2.1 | | | Interim, SAC |
| 2.5 | Listing of Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition | Intent-to-<br>Treat | 2.1 | | | Interim, SAC |
| 2.6 | Listing of WHO Functional Class Data | Intent-to-<br>Treat | 2.6 | | | Interim, SAC |
| 2.7 | Listing of Plasma NT-Pro BNP Concentration (ng/L) | Intent-to-<br>Treat | 2.7 | | | Interim, SAC |
| 2.8 | Listing of Exploratory Echocardiogram | Intent-to-<br>Treat | 2.8 | | | Interim, SAC |
| 2.9 | Listing of Cardiopulmonary Hemodynamics | Intent-to-<br>Treat | 2.9 | | | Interim, SAC |
| 2.10 | Listing of School Days | Intent-to-<br>Treat | 2.10 | | | Interim, SAC |
| 2.11 | Listing of Subject Global Assessment (SF10 Health Survey for Children) | Intent-to-<br>Treat | 2.11 | | | Interim, SAC |

# Safety Listings

| Listing<br>Number | Title | Population | Template<br>Listing | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
|---|---|---|---|---|---|---|
| 3.1 | Listing of Exposure and Compliance to Investigational Product | Safety | 3.1 | | | Interim, SAC |
| 3.2 | Listing of All Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.3 | Listing of Relationship between Adverse Event System Organ Class, Preferred Term and Verbatim Text | Safety | 3.3 | | | Interim, SAC |
| 3.4 | Listing of Subject Numbers for Specified Adverse<br>Events | Safety | 3.4 | | | Interim, SAC |
| 3.5 | Listing of Serious Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.6 | Listing of Fatal Serious Adverse Events | Safety | 3.2 | | | Interim, SAC |
| 3.7 | Listing of Adverse Events Leading to Permanent<br>Discontinuation of Study Treatment or Withdrawal<br>from Study | Safety | 3.2 | | | Interim, SAC |
| 3.8 | Listing of Haematology | Safety | 3.8 | | | Interim, SAC |
| 3.9 | Listing of Haematology Data for Subjects with<br>Abnormalities of Potential Clinical Concern | Safety | 3.9 | | | Interim, SAC |

| RAP | CONFIL | ENTIAL | | | | AMB1145 |
|---|---|---|---|---|---|---|
| | / | | | | | |
| Listing<br>Number | Title | Population | Template<br>Listing | Japanese<br>subgroup<br>analysis | Age<br>strata<br>subgroup<br>analysis | Deliverable |
| 3.10 | Listing of Clinical Chemistry | Safety | 3.8 | | | Interim, SAC |
| 3.11 | Listing of Clinical Chemistry Data for Subjects with Abnormalities of Potential Clinical Concern | Safety | 3.9 | | | Interim, SAC |
| 3.12 | Listing of Endocrinology Laboratory Data - Females only | Safety | 3.8 | | ADDED:<br>Footnote<br>(See<br>listing<br>3.22) | Interim, SAC |
| 3.13 | Listing of Liver Event Results and Time of Event Relative to Treatment | Safety | 3.13 | | | Interim, SAC |
| 3.14 | Listing of patient specific information for liver events | Safety | 3.14 | | | Interim, SAC |
| 3.15 | Listing of Medical Conditions for Subjects with Liver Events on Treatment | Safety | 3.15 | | | Interim, SAC |
| 3.16 | Listing of Liver Biopsy Details | Safety | 3.16 | | | Interim, SAC |
| 3.17 | Listing of Liver Imaging Details | Safety | 3.17 | | | Interim, SAC |
| 3.18 | Listing of Vital Signs | Safety | 3.18 | | | Interim, SAC |
| 3.19 | Listing of Vital Signs Data for Subjects with<br>Abnormalities of Potential Clinical Concern | Safety | 3.9 | | | Interim, SAC |
| 3.20 | Listing of Physical Examination | Safety | 3.20 | | | Interim, SAC |
| 3.21 | Listing of 12-Lead ECG Findings | Safety | 3.21 | | | Interim, SAC |
| 3.22 | Listing of Endocrinology Assessments | Safety | 3.22 | | ADDED:<br>Footnote | Interim, SAC |
| 3.23 | Listing of Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to tolerability issues | Safety | 2.1 | | | Interim, SAC |
| 3.24 | Listing of Pregnancy Results | Safety | 3.24 | | | Interim, SAC |
| 3.25 | Listing of Endocrinology Parameters - 20 Year Visit | Safety | 3.25 | | ADDED: Footnote | New Listing<br>for SAC |
| ovid-19 I | istings | | | | | |
| 3.26 | Listing of Country Level Start Dates of COVID-19 Pandemic Measures | Intent-to-<br>Treat | 3.26 | | | SAC |
| 3.27 | Listing of Visits and Assessments Impacted by COVID-19 Pandemic | Intent-to-<br>Treat | 3.27 | | | SAC |
| 3.28 | Listing of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | Safety | | | | SAC |

# 19.1.3. Figures

Efficacy Figures

| ITTICACY I | rgures / | | | | | |
|---|---|---|---|---|---|---|
| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age strata subgroup analysis | Deliverable |
| 2.1 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to Death (All Cause) | Intent-to-Treat | 3.1 | | | Interim, SAC |
| 2.2 | Box plots of 6 Minute Walking Distance (meters) by Visit | Intent-to-Treat | 3.4 | | | Interim, SAC |
| 2.3 | Box plots of Change from Baseline in 6 Minute Walking Distance (meters) by Visit | Intent-to-Treat | 3.4 | | | Interim, SAC |
| 2.4 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Clinical Worsening of PAH | Intent-to-Treat | 3.1 | | | Interim, SAC |
| 2,5 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to the addition of another targeted PAH therapeutic agent (prostanoids, PDE-5 inhibitors) | Intent-to-Treat | 3.1 | | | Interim, SAC |
| .6 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition | Intent-to-Treat | 3.1 | | | Interim, SAC |
| . 7 | Box plots of Plasma NT-Pro BNP concentration by Visit | Intent-to-Treat | 3.4 | | | Interim, SAC |
| 2.8 | Box plots of Change from Baseline in Plasma NT-Pro BNP concentration by Visit | Intent-to-Treat | 3.4 | | | Interim, SAC |
| 2.9 | Box plots of Exploratory Echocardiogram Data by Visit | Intent-to-Treat | 3.4 | X (Line plots of Exploratory Echocardiogra m Data by Subject) see template 3.11) | | Interim, SAC |
| 2.10 | Box plots of Change from Baseline in Exploratory Echocardiogram Data by Visit | Intent-to-Treat | 3.4 | | | Interim, SAC |

Safety Figures

| Figure<br>Number | Title | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age strata Deliverable subgroup analysis |
|---|---|---|---|---|---|
| 3.1 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Treatment-Emergent Adverse Event | Safety | 3.1 | | Interim, SAC |
| 3.2 | Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Serious Adverse Event | Safety | 3.1 | | Interim, SAC |
| 3.3 | Bar Chart of Treatment-Emergent Adverse Events Occurring in Two or More<br>Subjects in any Treatment Group | Safety | 3.3 | | Interim, SAC |
| 3.4 | Box plots of Haematology Data by Visit (Selected Parameters) | Safety | 3.4 | | Interim, SAC |

|---|---|---|---|---|---|---|---|
| Figure<br>Number | Title | | Population | Template<br>Figure | Japanese<br>subgroup<br>analysis | Age strata<br>subgroup<br>analysis | Deliverable |
| .5 | Box plots of Change from Baselin Parameters) | e in Haematology Data by Visit (Selected | Safety | 3.4 | | | Interim, SAC |
| .6 | Box plots of Chemistry Data by V | isit (Selected Parameters) | Safety | 3.4 | | | Interim, SAC |
| .7 | Box plots of Change from Baselin Parameters) | e in Chemistry Data by Visit (Selected | Safety | 3.4 | | | Interim, SAC |
| .8 | Patient Profiles of Liver Functi | on Tests | Safety | 3.8 | | | Interim, SAC |
| .9 | Box plots of Vital Signs Data by | Visit | Safety | 3.4 | | | Interim, SAC |
| .10 | Box plots of Change from Baselin | e in Vital Signs Data by Visit | Safety | 3.4 | | | Interim, SAC |
| .11 | Line plots of Endocrinology Asse | ssments by subject | Safety | 3.11 | | ADDED:<br>Footnote | Interim, SAC |
| .12 | Kaplan-Meier Survival Curves wit in dose of ambrisentan or other (prostanoids, PDE-5 inhibitors) | | Safety | 3.1 | | | Interim, SAC |


# 19.2. Data Display Specifications


Population: Intent-to-Treat

Table 1.1: Summary of Subject Disposition

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Subject status | | | | | |
| Completed | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Withdrawn | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Died | 1111 (0) | ( 0 ) | 1111 (0) | 1111 (0) | 1111 (0) |
| Died due to Covid-19 Complications | | | | | |
| Primary reason for study withdrawal * | | | | | |
| Adverse event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Lack of Efficacy | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Protocol Deviation | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Subject reached protocol defined stopping criteria | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Study closed/terminated | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Lost to Follow-up | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Investigator discretion | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Withdrew consent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Number of subjects who returned for a pubertal assess | sment | | | | |
| at 20-years of age | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |

Note: \* Percentages are based on the number of subjects in the treatment group.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Denominator for each primary reason for withdrawal is number of subjects in the Intent-to-Treat population per treatment group.

Population: Randomised

Table 1.2: Summary of Study Populations

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Randomised | XXX | XXX | XXX | XXX | XXX |
| Safety Population | XXX (%) | XXX (%) | XXX (%) | XXX (%) | XXX (%) |
| Intention-to-Treat population | XXX (%) | XXX (%) | XXX (%) | XXX (%) | XXX (%) |

Note: The Safety Population is defined as all subjects who received at least 1 dose of study drug. Subjects are considered as belonging to the treatment group according to the highest dose received.

The Intention-to-Treat (ITT) Population will consist of all subjects who received at least 1 dose of study drug. belonging to their treatment group at the start of study AMB114588.

Subjects are considered as

USER ID: Directory/Program.sas Date Time

Programming notes: See notes above relating to denominators for percentages.

Protocol: AMB114588

Population: Intent-to-treat


Table 1.3: Summary of Subjects by Country and Centre

| Country | Centre ID | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| XXXXXXXX | All | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | XXXXXX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| XXXXXXXX | All | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | XXXXXX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| XXXXXXXX | All | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | XXXXXX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.4: Summary of Inclusion/Exclusion Criteria Deviations

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Any criteria deviations | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Inclusion | | | | | |
| I1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| I2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | |
| Exclusion | | | | | |
| E1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| E2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | |

Note: Please refer to numbering of inclusion and exclusion criteria in protocol.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Only present criteria where there is at least one (total) deviation. "Any criteria deviations" is the number of subjects who had at least one deviation.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisentan<br>2.5mg | Ambrisentan<br>5mg | Ambrisentan<br>7.5mg | Ambrisentan<br>10mg | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (11 11111) |
| The state of the s | | | | | |
| Age (yrs) ** | ****** | 171717 | ***** | 77777 | ***** |
| N | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| Age (yrs)** | | | | | |
| N | XXX | XXX | XXX | XXX | XX (%) |
| <8 years | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| 8 - 11 years | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| 12 - <18 years | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| >=18 years | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Sex | | | | | |
| N | XXX | XXX | XXX | XXX | XX (%) |
| Female | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Male | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* At start of study treatment in AMB112529

<sup>\*</sup> At entry to AMB114588

<sup>\$</sup> A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisen<br>2.5mg<br>(N=XXX | ſ | Ambrisen<br>5mg<br>(N=XXX | | Ambrisen<br>7.5mg<br>(N=XXX | 1 | Ambriser<br>10mg<br>(N=XXX | | Total<br>(N=XXX | |
|---|---|---|---|---|---|---|---|---|---|---|
| Child Bearing Potential (Females only) * | | | | | | | | | | |
| N | XXX | | XXX | | XXX | | XXX | | XXX | |
| Pre-menarcheal | XX | (응) | XX | (응) | XX | (응) | XX | (%) | XX | (응) |
| Sterile (of child bearing age) | | (응) | XX | (응) | XX | | XX | (응) | | (%) |
| Potentially able to bear children | XX | (%) | XX | (%) | XX | (%) | XX | (%) | XX | (%) |
| Ethnicity ** | | | | | | | | | | |
| N | XXX | | XXX | | XXX | | XXX | | XXX | |
| Hispanic/Latino | XX | (응) | XX | (응) | XX | (응) | XX | (%) | XX | (응) |
| Not Hispanic/Latino | XX | (응) | XX | (응) | XX | (응) | XX | (응) | XX | (%) |
| Geographic Ancestry **\$ | | | | | | | | | | |
| n | XXX | | XXX | | XXX | | XXX | | XXX | |
| African American/African Heritage | XX | (%) | XX | (응) | XX | (응) | XX | (%) | XX | (응) |
| American Indian or Alaskan Native | XX | (응) | XX | (응) | XX | (응) | XX | (%) | XX | (응) |
| Asian - Central/South Asian Heritage | XX | (%) | XX | (%) | XX | (왕) | XX | (%) | XX | (응) |
| Asian - East Asian Heritage | XX | (%) | XX | (%) | XX | (왕) | XX | (%) | XX | (응) |
| Asian - Japanese Heritage | XX | (%) | XX | (%) | XX | (왕) | XX | (%) | XX | (응) |
| Asian - South East Asian Heritage | XX | (%) | XX | (%) | XX | (%) | XX | (%) | XX | (왕) |
| Native Hawaiian or Other Pacific Islander | XX | (응) | XX | (%) | XX | (%) | XX | (응) | XX | (%) |
| White - Arabic/North African Heritage | XX | (응) | XX | (%) | XX | (%) | XX | (응) | XX | (%) |
| White - White/Caucasian/European Heritage | XX | (왕) | XX | (%) | XX | (%) | XX | (왕) | XX | (응) |

Note: \*\* At start of study treatment in AMB112529

<sup>\*</sup> At entry to AMB114588

<sup>\$</sup> A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Weight (kg)* | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| Weight (kg)* | | | | | |
| N | XXX | XXX | XXX | XXX | XX (%) |
| <20 kg | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| 20 - <35 kg | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| 35 - <50 kg | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| >=50 kg | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Aetiology of PAH Randomised Strata ** | | | | | |
| n | XXX | XXX | XXX | XXX | XX (%) |
| Idiopathic (IPAH) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Familial (FPAH) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Persistent PAH despite surgical repair | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Secondary to connective tissue disease | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* At start of study treatment in AMB112529

<sup>\*</sup> At entry to AMB114588

<sup>\$</sup> A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.5: Summary of Demographic and Baseline Characteristics

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Duration of PAH (days)** | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| PAH Therapy Use ** | | | | | |
| n | XXX | XXX | XXX | XXX | XX (%) |
| Ongoing PAH therapy at baseline | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Prior PAH therapy, not ongoing at baseline | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| No PAH therapy recorded | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* At start of study treatment in AMB112529

\* At entry to AMB114588

\$ A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


| Table 1.5: | Summary c | of Demographic | and Baseline | Characteristics |
|------------|-----------|----------------|--------------|-----------------|
| | | Ambrisentan | Ambrisentan | Ambrisentan |
| | | 2.5mg | 5mg | 7.5mg |

| WHO Functional Class ** XXX | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| ##O Functional Class ** N | | 2.5mg<br>(N=XXX) | 5mg<br>(N=XXX) | 7.5mg<br>(N=XXX) | 10mg<br>(N=XXX) | (N=XXX) |
| N | WHO Functional Class ** | (2. 2.2.2.2) | (=: ======) | (=======) | (=: =====) | |
| Class III | | XXX | XXX | XXX | XXX | XX (%) |
| WHO Functional Class * XX (%) XX (%) XX (%) XX (%) XX (%) N Class II Class III XXX (%) XX (%) XX (%) XX (%) XX (%) XX (%) XX (%) XX (%) Class III XX (%) XX (%) XX (%) XX (%) XX (%) XX (%) XX (%) 6 minute walk data (m)** XXX XX | Class II | XX (%) | XX (%) | XX (%) | XX (%) | |
| N | Class III | | XX (%) | XX (%) | | XX (%) |
| Class III | WHO Functional Class * | | | | | |
| Class III | N | XXX | XXX | XXX | XXX | XX (%) |
| Class III | Class II | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| N XXX | Class III | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Mean XX.X XX.X XX.XX XX | 6 minute walk data (m) ** | | | | | |
| SD XX.XX XX | N | XXX | XXX | XXX | XXX | XXX |
| Q1 XX.X X | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median XX.X < | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q3 XX.X < | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. XX XXX | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Max. XX XX XX XX XX XX XXX | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| 6 minute walk data (m)* N | Min. | XX | XX | XX | XX | XX |
| N XXX | Max. | XX | XX | XX | XX | XX |
| Mean XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX <td>6 minute walk data (m)*</td> <td></td> <td></td> <td></td> <td></td> <td></td> | 6 minute walk data (m)* | | | | | |
| SD XX.XX XX | N | XXX | XXX | XXX | XXX | XXX |
| Q1 XX.X < | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median XX.X < | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q3 | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. XX XX XX XX XX | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. XX XX XX XX XX | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Max. XX XX XX XX XX | | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* At start of study treatment in AMB112529

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

<sup>\*</sup> At entry to AMB114588

<sup>\$</sup> A subject may be represented in more than one geographic ancestry group.

Q1 = 1st quartile, Q3 = 3rd quartile.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.6: Summary of Past Medical Conditions

| Classification | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Any condition | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Classification 1 | | | | | |
| Any condition | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| etc | | | | | |
| Classification 2 | | | | | |
| Any condition | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| etc | | | | | |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: "Any condition" relates to the number and percentage of subjects who had at least one condition. Subjects may be counted more than once across classifications.

Produce table for data collected in AMB112529 for the subset of subjects who entered AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.8: Summary of Concomitant Medications

| ATC Level 1 Preferred Term | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Endocrine & Metabolic | | | | | |
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Fluticasone propionate | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Beclomethasone dipropionate | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Anti-infectives & immunologicals | | | | | |
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Amoxycillin | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Amoxycillin trihydrate | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Clamoxyl | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Cefacior | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Cefproxil | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: A medication may be included in more than one ATC level category and appear more than once. Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Medications will be sorted in descending order of total incidence across treatment groups for the ATC level 1 and in descending order of total incidence for the preferred term within each ATC level. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.9: Summary of Ongoing Background PAH Therapy at Entry Visit to AMB114588

By Drug Class and Preferred Term

| PAH Therapy | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| | $(N-\Lambda\Lambda\Lambda)$ | (IN-VVV) | (IV-XXX) | (N-XXX) | |
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| PDE5i (monotherapy) | | | | | |
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | |
| Prostanoid (monotherapy) | | | | | |
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | |
| PDE5i and prostanoid in combination | | | | | |
| Any medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 1 + Preferred Term 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Preferred Term 3 + Preferred Term 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: For Table 1.10, data will be presented at 6 months after entry into AMB114588 and then annually as well as the final visit.

Protocol: AMB114588

Population: Intent-to-Treat


Table 1.11: Summary of Compliance to Investigational Product since last visit

| Planned Relative Time | Compliance assessment | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan 7.5mg (N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total (N=XXX) |
|---|---|---|---|---|---|---|
| | compilation appearment | (11 11111) | (11 11111) | (11 11111) | (11 11111) | (11 11111) |
| Month 3 | n | XXX | XXX | XXX | XXX | XXX |
| | 0% compliant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >0% and < 80% | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >= 80% and <= 120% | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >120% compliant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Month 6 | n | XXX | XXX | XXX | XXX | XXX |
| | 0% compliant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >0% and < 80% | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >= 80% and <= 120% | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >120% compliant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | Etc | | | | | |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits and End of Study.

Protocol: AMB114588

Population: Intent-to-treat


Table 1.12: Summary of Investigational Product Compliance Overall

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Overall % of visits at which subject is compliant | XX | XX | XX | XX | XX |
| N | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: Q1 = 1<sup>st</sup> quartile, Q3 = 3<sup>rd</sup> quartile.

Compliant visits are those at which subjects are  $\geq 80\%$  and  $\leq 120\%$  compliant. Compliance is determined by the site.

At a subject level compliance = 100\* (the number of visits at which the subject was compliant)/(the sum of all study visits for the subject). At a treatment group level the overall compliance = 100\* (the total number of visits at which all subjects in that group were compliant)/(the sum of all study visits for all subjects in that group).

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Population: Intent-to-treat


Table 1.13: Summary of initial dose of ambrisentan at entry to AMB114588 and highest dose received during study

| | | Н | ighest Dose | | |
|--------------|-------|-----|-------------|------|-------|
| Initial Dose | 2.5mg | 5mg | 7.5mg | 10mg | Total |
| 2.5 mg | XX | XX | XX | XX | XX |
| 5 mg | XX | XX | XX | XX | XX |
| 7.5 mg | XX | XX | XX | XX | XX |
| 10 mg | XX | XX | XX | XX | XX |
| Total | XX | XX | XX | XX | XX |

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|
|-----|--------------|-----------|

Population: Intent-to-treat


Table 1.14: Summary of initial dose of ambrisentan at entry to AMB114588 and final dose at end of study or termination

| | | ] | Final Dose | | |
|--------------|-------|-----|------------|------|-------|
| Initial Dose | 2.5mg | 5mg | 7.5mg | 10mg | Total |
| 2.5 mg | XX | XX | XX | XX | XX |
| 5 mg | XX | XX | XX | XX | XX |
| 7.5 mg | XX | XX | XX | XX | XX |
| 10 mg | XX | XX | XX | XX | XX |
| Total | XX | XX | XX | XX | XX |

USER ID: Directory/Program.sas Date Time

| .P | CONFIDENTIAL | AMB114588 |
|----|--------------|-----------|
|----|--------------|-----------|

Population: Intent-to-Treat


Table 1.15: Summary of Important Protocol Deviation

| | Ambrisentan<br>2.5mg | Ambrisentan 5mg | Ambrisentan<br>7.5mg | Ambrisentan 10mg | Total |
|---|---|---|---|---|---|
| Protocol Deviation Category | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Any Deviation | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Eligibility criteria not met | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Not withdrawn after developing withdrawal criteria | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Prohibited medication or device | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Visit window | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Informed consent procedure | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Administer/dispense study medication | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Failure to report SAE, Pregnancy, or liver function abnormalities per | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| protocol | | | | | |
| Study blind/ unblind procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Study treatment supply procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Biological specimen sample procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Assessment procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Diary Card procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Equipment procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Randomization procedures | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| IP taken inappropriately | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Procedures/Assessments not performed per protocol | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Other | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588 

Diagnosis

Population: Intent-to-Treat

Table 1.19

Summary of COVID-19 Assessments for Subjects with Suspected, Probable or Confirmed COVID-19 Case

| Assessments | Treatment A (N=300) | Treatment B (N=300) |
|-----------------------------|---------------------|---------------------|
| COVID-19 Case Diagnosis [1] | 100 (33%) | 100 (33%) |
| Confirmed | 29 (10%) | 29 (10%) |
| Probable | 50 (17%) | 50 (17%) |
| Suspected | 21 (7%) | 21 (7%) |
| COVID-19 Test Performed [2] | | |
| n | 100 | 100 |
| No | 50 (50%) | 50 (50%) |
| Yes | 50 (50%) | 50 (50%) |
| Result of the COVID-19 Test | | |
| n | 50 | 50 |
| Negative | 10 (20%) | 10 (20%) |
| Positive | 30 (60%) | 30 (60%) |
| Indeterminate | 10 (20%) | 10 (20%) |

<sup>[1]</sup> COVID-19 Case Diagnosis is based on WHO Definition as of dd-mmm-yyyy.

Programmer Notes: For COVID-19 Test Performed, the small n is based on the number of subjects with a COVID-19 Case Diagnosis.

For Result of the COVID-19 Test, the small n is based on the COVID-19 Test Performed=Yes. There are multiple collection forms, select the appropriate display format, PAN1 or PAN1A, depending on the form used in the study. Use PAN1 when the COVID-19 assessments can only be captured once during the study and use PAN1A if the COVID-19 assessments are captured using repeating form design.

<sup>[2]</sup> COVID-19 Test Performed is only captured for subjects with a COVID-19 Case Diagnosis.

Protocol: AMB114588 

Population: Intent-to-Treat

Table 1.20 Summary of Visits impacted by COVID-19 Pandemic

| | Treatment A | Treatment B | Total |
|---|---|---|---|
| | (N=100) | (N=100) | (N=200) |
| Any Visit Impacted | | | |
| Number of subjects with visits impacted | 80 (80%) | 80 (80%) | 160 (80% |
| | 00 (00%) | 00 (00%) | 100 (00% |
| Impact [4] | 25 (25%) | 25 (25%) | EO (2E) |
| MISSED VISIT | 25 (25%) | 25 (25%) | 50 (25% |
| Primary Reason for Impact [4] | 15 /150) | 15 /150\ | 20 (15) |
| SUBJECT ACQUIRED COVID-19 INFECTION [1] | 15 (15%) | 15 (15%) | 30 (15% |
| SUBJECT RELATED IMPACT [2] | 15 (15%) | 15 (15%) | 30 (15% |
| SITE RELATED IMPACT [3] | 15 (15%) | 15 (15%) | 30 (15% |
| SITE VISIT WITH ONE OR MORE ASSESSMENTS MISSED | 45 (45%) | 45 (45%) | 90 (45% |
| Primary Reason for Impact [4] | | | |
| SUBJECT ACQUIRED COVID-19 INFECTION [1] | 25 (25%) | 25 (25%) | 50 (25% |
| SUBJECT RELATED IMPACT [2] | 15 (15%) | 15 (15%) | 30 (15% |
| SITE RELATED IMPACT [3] | 15 (15%) | 15 (15%) | 30 (15% |
| REMOTE VISIT WITH NO ASSESSMENTS MISSED | 15 (15%) | 15 (15%) | 30 (15% |
| Primary Reason for Impact [4] | | | |
| SUBJECT ACQUIRED COVID-19 INFECTION [1] | 10 (10%) | 10 (10%) | 20 (10% |
| SUBJECT RELATED IMPACT [2] | 10 (10%) | 10 (10%) | 20 (10% |
| SITE RELATED IMPACT [3] | 10 (10%) | 10 (10%) | 20 (10% |
| REMOTE VISIT WITH ONE OR MORE ASSESSMENTS MISSED | 15 (15%) | 15 (15%) | 30 (15% |
| Primary Reason for Impact [4] | | | |
| SUBJECT ACQUIRED COVID-19 INFECTION [1] | 10 (10%) | 10 (10%) | 20 (10% |
| SUBJECT RELATED IMPACT [2] | 10 (10%) | 10 (10%) | 20 (10% |
| SITE RELATED IMPACT [3] | 10 (10%) | 10 (10%) | 20 (10% |
| Visit # | | | |
| Number of impacted subjects at the visit (n) | 60 | 60 | 120 |
| Impact | | | |
| MISSED VISIT | 6 (10%) | 6 (10%) | 12 (10% |
| Primary Reason for Impact | | | |
| SUBJECT ACQUIRED COVID-19 INFECTION [1] | 3 (5%) | 3 (5%) | 6 (5% |
| SUBJECT RELATED IMPACT [2] | 0 | 0 | 0 |
| SITE RELATED IMPACT [3] | 3 (5%) | 3 (5%) | 6 (5% |
| SITE VISIT WITH ONE OR MORE ASSESSMENTS MISSED | 36 (60%) | 36 (60%) | 72 (60% |
| Primary Reason for Impact | | | |
| SUBJECT ACQUIRED COVID-19 INFECTION [1] | 0 | 0 | 0 |

|----------------------------|--------------|-------------|-----------|
| SUBJECT RELATED IMPACT [2] | 6 (10%) | 6 (10%) 12 | 2 (10%) |
| SITE RELATED IMPACT [3] | 30 (50%) | 30 (50%) 60 | (50%) |

Visit ...

- [1] Subject acquired COVID-19 includes suspected, probable and confirmed.
- [2] Subject related impact include subject discretion and travel restrictions.
- [3] Site related impacts include site temporarily closed, site staff unavailable, and study drug unavailable.
- [4] Subjects may be counted in more than one category.

/Directory/program.sas 01JAN2002 12:01

Programmer notes: After the overall summary of any impacted visits, the summary is then produced by visit starting with the first impacted visit. This is represented in the mock-up as # for the first impacted visits and #+1 for each visit thereafter.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.1: Summary of Time to Death (All cause) (days)

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| N | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.2: Summary of 6 Minute Walking Distance (meters)

| Treatment | Planned | n | Mean | SD | Q1 | Median | Q3 | Min. | Max |
|---|---|---|---|---|---|---|---|---|---|
| | Relative Time | | | | | | | | |
| Ambrisentan | Baseline** | | | | | | | | |
| 2.5mg | Overall | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| 3 | With oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Without oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Entry Visit* | | | | | | | | |
| | Overall | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | With oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Without oxygen use | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 6 | | | | | | | | |
| | Etc | | | | | | | | |
| Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| Ambrisentan<br>7.5mg<br>(N=XXX) | Etc | | | | | | | | |
| Ambrisentan<br>10mg<br>(N=XXX) | Etc | | | | | | | | |
| Total (N=XXX) | Etc | | | | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.5: Summary of Walking Duration (minutes) for subjects who walked less than six minutes

| Treatment | Number of subjects who attempted the 6 minute walk | | n | Mea | an | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan 2.5mg | XX | Baseline** | XX (§ | ;) XX | Х.Х | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | XX<br>XX<br>XX | Entry Visit* Month 6 Etc | XX (9<br>XX (9<br>XX (9 | ) XX | X.X<br>X.X | XX.XX<br>XX.XX<br>XX.XX | XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X | XX<br>XX<br>XX | XX<br>XX<br>XX |
| Ambrisentan<br>5mg<br>(N=XXX) | | Etc | | | | | | | | | |
| Ambrisentan<br>7.5mg<br>(N=XXX) | | Etc | | | | | | | | | |
| Ambrisentan<br>10mg<br>(N=XXX) | | Etc | | | | | | | | | |
| Total<br>(N=XXX) | | Etc | | | | | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.6: Summary of use of Oxygen during 6 Minute Walking exercise (L/min)

| Treatment | Number of subjects who attempted the 6 minute walk | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan 2.5mg | XX | Baseline** | XX (%) | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | XX<br>XX<br>XX | Entry Visit* Month 6 Etc | XX (%)<br>XX (%)<br>XX (%) | XX.X | XX.XX<br>XX.XX<br>XX.XX | XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X | XX<br>XX<br>XX | XX<br>XX<br>XX |
| Ambrisentan<br>5mg<br>(N=XXX) | | Etc | | | | | | | | |
| Ambrisentan 7.5mg (N=XXX) | | Etc | | | | | | | | |
| Ambrisentan<br>10mg<br>(N=XXX) | | Etc | | | | | | | | |
| Total<br>(N=XXX) | | Etc | | | | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.7: Summary of Time to the first Clinical Worsening of PAH (days)

| | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|--------|-------------|-------------|-------------|-------------|-----------|
| | 2.5mg | 5mg | 7.5mg | 10mg | (N=XXX) |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| N | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.8: Summary of Clinical Worsening of PAH

| | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Subjects with at least one criteria | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Death (all cause) or placed on active list for lung transplant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Hospitalisation for worsening of PAH | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Addition/increased dose of other targeted PAH therapetic agents and/or atrial septostomy | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| PAH related deterioration | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| PAH related deterioration:- | | | | | |
| Increase from baseline in WHO functional class | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Deterioration in exercise testing | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Clinical signs or symptoms of right sided heart failure | XX (%) | XX (%) | XX (%) | XX (%) | XX (응) |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

|-----|--------------|-----------|

Population: Intent-to-Treat

Table 2.9: Summary of Time to the addition of another targeted PAH therapeutic agent (prostanoids, PDE-5 inhibitors) (days)


| | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|
| | 2.5mg | 5mg | 7.5mg | 10mg | (N=XXX) |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| ue to Deterioration of Clinical | | | | | |
| ondition | | | | | |
| N | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| revious therapy | | | | | |
| N | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean<br>SD | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX | XX.X<br>XX.XX |
| Mean<br>SD<br>Q1 | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X |
| Mean<br>SD<br>Q1<br>Median | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X |
| Mean<br>SD<br>Q1<br>Median<br>Q3 | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |
| Mean<br>SD<br>Q1<br>Median | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X |
| Mean<br>SD<br>Q1<br>Median<br>Q3 | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |
| Mean SD Q1 Median Q3 Min. | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |
| Mean SD Q1 Median Q3 Min. Max. | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |
| Mean SD Q1 Median Q3 Min. Max. | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |

Note: Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Use CONMEDS dataset where CMTYPCD is 84(PAH Therapy) and CMSTRSCD = 46 (Deterioration of clinical condition) or = 47 (Lack of beneficial effect with previous therapy).

Population: Intent-to-Treat


Table 2.10: Summary of Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition (days)

| | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|
| | 2.5mg | 5mg | 7.5mg | 10mg | (N=XXX) |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| N | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Use CONMEDS dataset where CMTYPCD is 84(PAH Therapy) and CMSTRSCD = 46 (Deterioration of clinical condition) or EXPOSURE dataset where EXCHRSCD = 58 (Deterioration of clinical condition).

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.11: Summary of WHO Functional Class

| Treatment | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan<br>2.5mg | Baseline** | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Entry Visit* Month 6 | XX<br>XX | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | XX | XX |
| Ambrisentan<br>5mg<br>(N=XXX) | Etc | XX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan 7.5mg (N=XXX) | Etc | | | | | | | | |
| Ambrisentan<br>10mg<br>(N=XXX) | Etc | | | | | | | | |
| Total<br>(N=XXX) | Etc | | | | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

There are 4 grades of WHO FC based on symptom severity (Grades mapped to numeric scale 1-4 (i.e. Class IV=4).

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Table 2.13: Summary of WHO Functional Class Shifts from Baseline by Visit

| | Planned<br>Relative | WHO<br>Functional | Baseline**<br>WHO Functional Class | |
|---|---|---|---|---|
| Treatment | Time | Class _ | II | III |
| Ambrisentan 2.5mg (N=XXX) | Entry Visit* | I | XX (%) | XX (%) |
| - | - | II | XX (%) | XX (%) |
| | | III | XX (%) | XX (%) |
| | | IV | XX (%) | XX (%) |
| | | Unknown/ | XX | XX |
| | | Not Recorded | | |
| | Month 6 | I | XX (%) | XX (%) |
| | | II | XX (%) | XX (%) |
| | | III | XX (%) | XX (%) |
| | | IV | XX (%) | XX (%) |
| | | Unknown/ | XX | XX |
| | | Not Recorded | | |
| | Etc | | | |
| Ambrisentan 5mg (N=XXX) | Etc | | | |
| Ambrisentan 7.5mg (N=XXX) | Etc | | | |
| Ambrisentan 10mg (N=XXX) | Etc | | | |
| Total (N=XXX) | Etc | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

There are 4 grades of WHO FC based on symptom severity (

Grades mapped to numeric scale 1-4 (i.e. Class IV=4).

Baseline WHO functional class not shown for III and IV because no subjects met the criteria for these categories at baseline.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.14: Summary of WHO Functional Class Change from Baseline Categorisation

| Planned Relative Time | WHO Category | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Entry Visit* | N | XXX | XXX | XXX | XXX | XXX |
| | Improved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | No Change | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Deteriorated | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | <b>-</b> 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | -1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | 0 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | +1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | +2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

There are 4 grades of WHO FC based on symptom severity (CCI Grades mapped to numeric scale 1-4 (i.e. Class IV=4).

Change categorisation (based on -2, -1, 0, +1, +2);

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.15: Summary of plasma NT-Pro BNP concentration (ng/L)

| Treatment | Planned | n | Geometric | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| | Relative Time | | Mean | [logs] | | | | | |
| Ambrisentan<br>2.5mg | Baseline** | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Entry Visit* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 6 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Etc | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| Ambrisentan | Etc | | | | | | | | |

Ambrisentan Etc..

10mg (N=XXX)

7.5mg (N=XXX)

Total Etc.. (N=XXX)

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|

Population: Intent-to-Treat


Table 2.17: Summary of Exploratory Echocardiogram

| Planned | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| Relative Time | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Baseline** | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Pericardial | N | XXX | XXX | XXX | XXX | XXX |
| Effusion | Absent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Trace: separation of pericardial layers in both systole and diastole | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Small: diastolic separation equals 1cm | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Moderate: diastolic separation of 1 to 2cm | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Large: diastolic separation equals 2cm | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Mean right | N | XXX | XXX | XXX | XXX | XXX |
| Atrial | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Pressure | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| - | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Tricuspid | N | XXX | XXX | XXX | XXX | XXX |
| Annular | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Plane | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Systolic | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Excursion | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| (cm) | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits (including Entry Visit), End of Study and Follow-Up.

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

Population: Intent-to-Treat


Table 2.17: Summary of Exploratory Echocardiogram

| Planned | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| Relative Time | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Baseline** | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Eccentricity | N | XXX | XXX | XXX | XXX | XXX |
| Index | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Systolic / | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Eccentricity | N | XXX | XXX | XXX | XXX | XXX |
| Index | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Diastolic | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits (including Entry Visit), End of Study and Follow-Up.

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Population: Intent-to-Treat


Table 2.17: Summary of Exploratory Echocardiogram

| Planned | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| Relative Time | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Baseline** | | (N=XXX) | (N=XXX) | (N=XXX) | Ambrisentan 10mg (N=XXX) XXX XX.X XX.X XX.X XX.X XX.X XX.X | (N=XXX) |
| | / | | | | | |
| Tricuspid | N | XXX | XXX | XXX | | XXX |
| Regurgitant | Mean | XX.X | XX.X | XX.X | | XX.X |
| Jet Velocity / | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| (m/s) | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Right | N | XXX | XXX | XXX | XXX | XXX |
| entricular/ | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| ressure | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits (including Entry Visit), End of Study and Follow-Up.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.18: Summary of Change from Baseline in Exploratory Echocardiogram

| Planned Relati | ve / | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| Time | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Entry Visit* | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Pericardial | n | XXX | XXX | XXX | XXX | XXX |
| Effusion | No Change | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Absent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Improved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Worsened | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Mean right | n | XXX | XXX | XXX | XXX | XXX |
| Atrial | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Pressure | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Tricuspid | n | XXX | XXX | XXX | XXX | XXX |
| Annular | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Plane | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Systolic | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Excursion | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| (cm) | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.18: Summary of Change from Baseline in Exploratory Echocardiogram

| Planned | / | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| Relative Time | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Entry Visit* | | (N=XXX) | (N=XXX) | (N=XXX) | 10mg (N=XXX) XXX | (N=XXX) |
| Eccentricity | n | XXX | XXX | XXX | XXX | XXX |
| Index / | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Systolic | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Eccentricity | N | XXX | XXX | XXX | XXX | XXX |
| Index | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Diastolic | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time
Protocol: AMB114588

Population: Intent-to-Treat


Table 2.18: Summary of Change from Baseline in Exploratory Echocardiogram

| Planned Relativ<br>Time<br>Entry Visit* | е | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Tricuspid | N | XXX | XXX | XXX | XXX | XXX |
| Regurgitant / | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Jet Velocity | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| (m/s) | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Right | N | XXX | XXX | XXX | XXX | XXX |
| Ventricular | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| Pressure | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| (mmHg) | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up.

Protocol: AMB114588

Population: Intent-to-treat


Table 2.19: Summary of Number of Subjects with School Days

| Planned Relative Time | | isentan<br>.5mg | | risentan<br>5mg | | risentan<br>'.5mg | | isentan<br>10mg | 7 | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | (1 | N=XX) | (1 | N=XX) | ( | N=XX) | (1 | A=XX) | ( | N=XX) |
| Baseline** | | | | | | | | | | |
| Subjects with scheduled days | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Subjects with at least one scheduled day missed | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Number of scheduled days missed / | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) |
| Number of scheduled days | | | | | | | | | | |
| Subjects with at least one scheduled day missed due to PAH | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Number of scheduled days missed due to PAH / | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Number of scheduled days | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) |
| Entry Visit* | | | | | | | | | | |
| Subjects with scheduled days | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Subjects with at least one scheduled day missed | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Number of scheduled days missed /<br>Number of scheduled days | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) |
| Subjects with at least one scheduled day missed due to PAH | xx | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Number of scheduled days missed due to PAH / | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Number of scheduled days | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) | xx/xxx | (xx%) |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

This summary excludes subjects with 0 scheduled days of school for the given period.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.20: Summary Statistics of School Days

| Planned Relative Time | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Baseline** | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Number | N | XXX | XXX | XXX | XXX | XXX |
| of scheduled days | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Number | N | XXX | XXX | XXX | XXX | XXX |
| of missed days | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Number | N | XXX | XXX | XXX | XXX | XXX |
| of missed days | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| due to PAH | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

This summary excludes subjects with 0 scheduled days of school for the given period.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.20: Summary Statistics of School Days

| Planned Relative Time | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Entry Visit | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Proportion of days | n | XXX | XXX | XXX | XXX | XXX |
| missed (%) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Proportion of days | N | XXX | XXX | XXX | XXX | XXX |
| missed due to PAH(%) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

This summary excludes subjects with 0 scheduled days of school for the given period.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Table 2.22: Summary of Subject Global Assessment (SF10 Health Survey for Children)

| Planned Relative Time | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| | | 2.5mg | 5mg | 7.5mg | 10mg | |
| Baseline** | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Physical Health Summary | n | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Psychosocial Summary | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat

Table 2.24: Summary of SF10 Health Survey - Number and Percentage of Subjects with Particular Item Responses


| Planned Relative Time | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|
| | 2.5mg | 5mg | 7.5mg | 10mg | |
| Baseline** | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Completed SF-10 ^ | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| In general, would you say your child's health is | | | | | |
| N | XX | XX | XX | XX | XX |
| Excellent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Very Good | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Good | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Fair | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Poor | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| During the past 4 weeks, has your child been limited | | | | | |
| doing things that take some energy such as riding a | | | | | |
| bike or skating due to HEALTH problems? | | | | | |
| N | XX | XX | XX | XX | XX |
| Yes, limited a lot | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Yes, limited some | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Yes, limited a little | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| No, not limited | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| During the past 4 weeks, has your child been limited | | | | | |
| during bending, lifting or stooping due to HEALTH | | | | | |
| problems? | | | | | |
| N | XX | XX | XX | XX | XX |
| Yes, limited a lot | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Yes, limited some | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Yes, limited a little | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| No, not limited | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| etc | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

<sup>\*</sup> Entry Visit is at entry to AMB114588.

<sup>^</sup> Completed at least one of the 10 items of SF-10

|-----|--------------|-----------|
|-----|--------------|-----------|

Protocol: AMB114588 

Population: Intent-to-treat

Table 2.25

Number of subjects who achieved an increase in 6MWD >=20 metres

| | N=XX |
|----------------------------------------------------------|----------|
| >/= 20 meters increase from baseline (LOCF) at 12 months | xx (xx%) |
| >/= 20 meters increase from baseline at last observation | xx (xx%) |

Note: Baseline is the last value recorded prior to the start of study treatment from AMB112529. USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|

Protocol: AMB114588

Population: Intent-to-treat

Table 2.26

Number of subjects who achieved an increase in 6MWD >=20 metres by Idiopathic group

| Idiopathic group | | N=100 |
|---|---|---|
| Idiopathic group | <pre>&gt;/= 20 meters increase from baseline at 12 months (LOCF) &gt;/= 20 meters increase from baseline at last observation</pre> | xx (xx%)<br>xx (xx%) |
| Non-idiopathic group | <pre>&gt;/= 20 meters increase from baseline at 12 months (LOCF) &gt;/= 20 meters increase from baseline at last observation</pre> | xx<br>xx (xx%)<br>xx (xx%) |


Note: Baseline is the last value recorded prior to the start of study treatment from AMB112529.

'Idiopathic group' refers to those with an idiopathic aetiology of PAH in 112529, and 'non-idiopathic' refers to those classified as having: an aetiology of familial, persistent PAH despite surgical repair, or secondary to connective tissue disease.

For subjects with missing data at 12 months, the post-baseline last observation was carried forward (LOCF) to the 12 month visit.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588


Population: Intent-to-treat

Table 2.27

Number of subjects who achieved an NT-proBNP level of less than 1200  $\mbox{ng/L}$ 

NT-proBNP level of less than 1200 ng/L at 12 months (LOCF)

NT-proBNP level of less than 1200 ng/L at last observation

xx (xx%)

xx (xx%)

Note: For subjects with missing data at 12 months, the post-baseline last observation was carried forward (LOCF) to the 12 month visit.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588


Population: Intent-to-treat

Table 2.28

Number of subjects who achieved an NT-proBNP level of less than 1200 ng/L by Idiopathic group

| Idiopathic group | | N=xx |
|---|---|---|
| Idiopathic group | NT-proBNP level of less than 1200 ng/L at 12 months (LOCF) NT-proBNP level of less than 1200 ng/L at last observation | xx (xx%)<br>xx (xx%) |
| Non-idiopathic group | NT-proBNP level of less than 1200 ng/L at 12 months (LOCF) | xx (xx%) |
| | NT-proBNP level of less than 1200 ng/L at last observation | xx (xx%) |

Note: 'Idiopathic group' refers to those with an idiopathic aetiology of PAH in 112529, and 'non-idiopathic' refers to those classified as having: an aetiology of familial, persistent PAH despite surgical repair, or secondary to connective tissue disease.

For subjects with missing data at 12 months, the post-baseline last observation was carried forward (LOCF) to the 12 month visit.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588 

Population: Intent-to-treat

Table 2.29
Distribution of NT-proBNP levels at baseline and extent of change during treatment

NT-proBNP value above 1200 ng/L at baseline x (18%) How many stayed over 1200 x (3%) How many had at least 1 value < 1200 x (13%) x (13%) How many had value <1200 as last value Other (a) x (3%) NT-proBNP value above 1200 ng/L at any time during the study xx (29%) NT-proBNP value between 500 ng/L and 1200 ng/L at baseline x (8%) How many had at least 1 value >1200? x (3%) and how many of these stayed over 1200? x (3%) How many stayed between 500 and 1200? x (3%) How many fell below 500 x (5%) Of those how many were <500 as last value? x (3%) Other (b) x (3%) NT-proBNP value < 500 ng/L at baseline xx (71%) How many had at least 1 value > 1200 x (8%) and of these how many stayed over 1200? x (5%) Other (c) x (3%)

| Note | | |
|------|---------|---------------------------------------------|
| (a) | Subject | did not have a baseline visit in AMB112529. |
| (b) | Subject | only had a baseline value. |
| (C) | Subject | went up to>1200, back down to 500-1200 |
| (d) | Subject | fell below 500 then up above 1200 |
| (e) | Subject | went up to 500-1200 but ended above 1200 |
| (f) | Subject | fell below 500 then back up to 500-1200 |

how many stayed there?

How many stayed below 500?

How many rose to between 500 and 1200?

USER ID: Directory/Program.sas Date Time

Other (d)

x (13%)

x (5%)

x (8%)

xx (55%)

Page 1 of 2

Protocol: AMB114588

Population: Intent-to-treat

## Table 2.30

Distribution of NT-proBNP levels at baseline and extent of change during treatment - by Idiopathic group

Group: Idiopathic group

| | N=x | ΧX |
|---|---|---|
| Idiopathic group | xx | |
| NT-proBNP value above 1200 ng/L at baseline How many stayed over 1200 How many had at least 1 value < 1200 How many had value <1200 as last value Other (a) | X<br>XX<br>XX | <pre>&lt; (xx%) (x%) &lt; (xx%) &lt; (xx%) &lt; (x%)</pre> |
| NT-proBNP value above 1200 ng/L at any time during the study | xx | (xx%) |
| NT-proBNP value between 500 ng/L and 1200 ng/L at baseline How many had at least 1 value >1200? | x<br>0 | (xx%) |
| and how many of these stayed over 1200? | | (x%) |
| How many stayed between 500 and 1200? | | (x%) |
| How many fell below 500 | | (x%) |
| Of those how many were <500 as last value? | X | (x%) |
| NT-proBNP value < 500 ng/L at baseline | XX | (63%) |
| How many had at least 1 value > 1200 | X | (x%) |
| and of these how many stayed over 1200? | X | (x%) |
| Other (b) | X | (x%) |
| How many rose to between 500 and 1200? | X | (x%) |
| how many stayed there? | X | (x%) |
| Other (c) | X | (x%) |
| How many stayed below 500? | XX | (x%) |

## Group: Non-idiopathic group-all other categories

| | N=x: | X<br> |
|--------------------------------------------------------------|------|-------|
| Number in non-idiopathic group | XX | |
| NT-proBNP value above 1200 ng/L at baseline | 0 | |
| How many stayed over 1200 | 0 | |
| How many had at least 1 value $<$ 1200 | 0 | |
| How many had value <1200 as last value | 0 | |
| NT-proBNP value above 1200 ng/L at any time during the study | х | (xx%) |
| NT-proBNP value between 500 ng/L and 1200 ng/L at baseline | X | (xx%) |
| How many had at least 1 value >1200? | X | (xx%) |
| and how many of these stayed over 1200? | X | (xx%) |
| How many stayed between 500 and 1200? | X | |
| How many fell below 500 | X | (xx%) |
| Of those how many were <500 as last value? | X | (xx%) |
| Other (d) | X | (xx%) |
| NT-proBNP value < 500 ng/L at baseline | XX | (xx%) |
| How many had at least 1 value > 1200 | 0 | . , |

|---------------------------------------|--------------|-----------|
| and of these how many stayed over | 1200? | 0 |
| How many rose to between 500 and 1200 | 0? | x (xx%) |
| how many stayed there? | | x (xx%) |
| Other (e) | | x (xx%) |
| How many stayed below 500? | | 0 (xx%) |

## Note:

(a) Subject
(b) Subject
(c) Subject
(d) Subject
(d) Subject
(e) Subject
(f) Subject
(f) Subject
(f) Subject
(f) Subject
(g) Subject
(g) Su

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|
|-----|--------------|-----------|

Protocol: AMB114588 

Population: Intent-to-Treat

Table 2.31

The Event Rate of the Clinical Worsening Endpoint per 100 Patient-Years

| Treatment | N | The number of subjects with at least one clinical worsening | Total exposure time (year) | Event rate per 100 patient-years |
|---|---|---|---|---|
| Total | хх | xx | XXXX.X | X.X |

Note: Total Exposure time in years is calculated by the sum for all subjects of (last exposure date - first exposure date + 1) / 365.25. If the last exposure date is missing, the last study visit date is used.

For the subjects with at least one clinical worsening, the first event date should be used instead of the last exposure date.

Event rate per 100 patient-years: The number of subjects with at least one clinical worsening / Total exposure time (year) \* 100;

Protocol: AMB114588 Population: Safety


Table 3.1: Summary of Exposure to Investigational Product

| | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| | | 2.5mg | 5mg | 7.5mg | 10mg | |
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Number of days | n | XXX | XXX | XXX | XXX | XXX |
| of exposure | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| <del>-</del> | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Interval of days | n | XXX | XXX | XXX | XXX | XXX |
| of exposure | <=1 month | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| - | >1 month to <=2 months | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | >2 month to <=3 months | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Etc | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: For each patient, exposure (days) = date of last dose of study drug - first dose date + 1 day.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

For subjects missing their last exposure date at the time of study end, their last visit date in the study was used.

Protocol: AMB114588 Population: Safety


Table 3.2: Summary of Treatment-Emergent Adverse Events

| System Organ Class Preferred term | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Gastrointestinal disorders | | | | | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dyspepsia | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nausea | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nervous system disorders | | | | | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Headache | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dizziness | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Somnolence | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Tremor | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Sedation | XX (%) | XX (%) | XX (%) | XX (%) | XX (% |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Events will be sorted in descending order of total incidence across treatment groups for the System Organ Class and in descending order of total incidence for the preferred term within each System Organ Class. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Protocol: AMB114588 Population: Safety


Table 3.3: Summary of Treatment-Emergent Adverse Events by Preferred Term

| Preferred term | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dyspepsia | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nausea | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Headache | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dizziness | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Somnolence | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Tremor | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Sedation | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Protocol: AMB114588 Population: Safety


Table 3.4: Summary of Treatment-Emergent Adverse Events by Maximum Intensity

| | | Ambrisenta: 2.5mg | n | | Ambrisentar<br>5mg | n | | Ambrisenta: 7.5mg | n | | Ambrisenta<br>10mg | ın |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | (N=XXX) | | | (N=XXX) | | | (N=XXX) | | | (N=XXX) | |
| | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| System Organ Class Preferred Term | | | | | | | | | | | | |
| Piereried leim | | | | | | | | | | | | |
| Any Event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Cardiovascular<br>disorders | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Any Event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Hypertension | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Syncope | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Aneurysms | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Hypotension Etc | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Repeat display for Total group on following page. Subjects who experience the same event several times, with different intensities/grades, will only be counted with the maximum intensity/grade. For example, a subject who had three headaches, two severe and one mild, is counted only once, under the preferred term "Headache" in the "Severe" column of the table. Likewise, each subject is counted only once, at the maximum severity/grade, within each SOC even though they may have several different PT events at different intensities/grades within that SOC. Events will be sorted in descending order of total incidence across treatment groups for the System Organ Class and in descending order of total incidence for the preferred term within each System Organ Class. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Protocol: AMB114588 Population: Safety


Table 3.5: Summary of Treatment-Emergent Adverse Events by Action Taken with IP

| System Organ Class<br>Preferred term<br>Action Taken | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| <system 1="" class="" organ=""></system> | | | | | |
| <any event=""></any> | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| IP withdrawn | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose interrupted | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose reduced | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose not changed | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose increased | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Not applicable | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| <preferred 1="" term=""></preferred> | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| IP withdrawn | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose interrupted | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose reduced | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose not changed | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dose increased | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Not applicable | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Subjects who experience the same event several times, with different Action Taken, will only be counted once for the overall and Preferred Term category, but more than once in the Action Taken categories. Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.


Population: Safety

Table 3.8: Summary of Cumulative Incidence of Treatment-Emergent Adverse Events by Time to First Occurrence

Treatment: Ambrisentan 2,5mg (N=XXX)

| | | | Time Sind | ce Start of St | udy Medication | n in AMB114588 | } | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred term | <=3<br>months | >3 to <=6 months | >6 to <=9 months | Etc | Etc | Etc | Etc | Overall |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Gastrointestinal | | | | | | | | |
| disorders | | | | | | | | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dyspepsia | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nausea | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Nervous system disorde | rs | | | | | | | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Headache | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Dizziness | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Somnolence | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Tremor | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Sedation | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order. Repeat for all Ambrisentan and Total groups.

Protocol: AMB114588 Population: Safety


Table 3.10: Summary of Serious Treatment-Emergent Adverse Events - Number of Subjects and Occurrences

| System Organ Class<br>Preferred Term | Treatment<br>Group | Subjects<br>Affected,<br>Number | Subjects<br>Exposed,<br>Number | Occurrences<br>All, Number | Occurrences<br>Causally<br>Related to<br>Treatment,<br>Number* | Fatalities,<br>Number | Fatalities Causally Related to Treatment, Number* |
|---|---|---|---|---|---|---|---|
| CARDIAC DISORDERS | | | | | | | |
| Atrial fibrillation | Ambrisentan<br>2.5mg | Х | Х | х | Х | х | Х |
| | Ambrisentan<br>5mg | х | Х | х | Х | х | х |
| | Ambrisentan<br>7.5mg | х | Х | х | Х | Х | Х |
| | Ambrisentan<br>10mg | Х | Х | x | Х | х | Х |
| | Total | X | Х | X | Х | X | X |

Bradyarrhythmia etc

Note: \* Drug-related as determined by the investigator.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|
|-----|--------------|-----------|

Protocol: AMB114588 Population: Safety


Table 3.11: Summary of Serious Treatment-Emergent Adverse Events by Outcome

| System Organ Class Preferred term Outcome | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan 7.5mg (N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| ouccome | , | , , | , , | , | |
| Any event | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| <system 1="" class="" organ=""></system> | | | | | |
| <any event=""></any> | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Recovering/Resolving | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved with sequelae | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Not Recovered/ Not Resolved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| <preferred 1="" term=""></preferred> | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Recovering/Resolving | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Recovered/Resolved with sequelae | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Not Recovered/ Not Resolved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Subjects who experience the same event several times, with different Outcome, will only be counted once for the overall and Preferred Term category, but more than once in the Outcome categories. Events will be sorted in descending order of total incidence across treatment groups for the preferred term. If the total incidence for any two or more preferred terms is equal, they will be presented in alphabetical order.

Protocol: AMB114588 Population: Safety

Central/Local Laboratory
Parameter: <Parameter (units)>


Table 3.21: Summary of Haematology Data

| Treatment | Planned<br>Relative Time | N | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Ambrisentan<br>2.5mg | Baseline** | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| (N=XXX) | Entry Visit* | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 1 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 2 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 3 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 4 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 5 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Month 6 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Etc | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| Ambrisentan | Etc | | | | | | | | |

5mg (N=XXX)

Ambrisentan Etc..

7.5mg (N=XXX)

Ambrisentan Etc..

10mg (N=XXX)

Total Etc..

(N=XXX)

Note:  $\star\star$  Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up. Absolute value tables done separately for central and local labs. Change from baseline required only for the subset of subjects who have QUEST Central labs throughout.


Population: Safety

Table 3.23: Summary of Haematology Data of Potential Clinical Concern

Central/Local Laboratory

Parameter: <Parameter (units) [Reference range = xx.x to xx.x ]>

| Planned<br>Relative Time | Category | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Baseline** | N | XXX | XXX | XXX | XXX | |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Intry Visit* | И | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Month 1 | И | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Month 2 | И | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | | |
| Any time<br>post-baseline | N | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | <pre>&lt; reference range low</pre> | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

For 'Any time in AMB114588 (Entry to End of Study)':-

Subjects with both Normal and Low values are counted once under their worst case (Low).

Subjects with both Normal and High values are counted once under their worst case (High).

Subjects with both High and Low values are counted under both categories.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up.

<sup>\*</sup> Entry Visit is at entry to AMB114588.

|-----|--------------|-----------|


Population: Safety

Table 3.29: Summary of Liver Events Assessment

| | Ambr | isentan | Ambr | isentan | Ambr | isentan | Ambr | isentan | T | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | 2 | .5mg | | 5mg | 7 | .5mg | 1 | L0mg | | |
| | (N | =XXX) | (N | =XXX) | (N | =XXX) | (N: | =XXX) | ( N | N=XXX) |
| Subjects reporting a significant liver chemistry result * | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |
| Subjects with event occurring while receiving study treatment | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |
| Subjects with event occurring after stopping study treatment | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |

Note: \* A significant liver chemistry result is any result which meets the stopping criteria defined in the protocol.

Detailed information on liver events assessment can be found in related listings.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588 Population: Safety


Table 3.30 Summary of Vital Signs

| Parameter | Treatment | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| <parameter (units)=""></parameter> | Ambrisentan<br>2.5mg | Baseline** | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Entry Visit | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | , | Month 3 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 6 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 9 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Etc | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| | Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| | Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| | Total<br>(N=XXX) | Etc | | | | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up. Include Height, Weight, Systolic BP, Diastolic BP, Heart Rate, BSA and BMI.

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.


Population: Safety

Table 3.32: Summary of Vital Signs Data of Potential Clinical Concern

Parameter: <Parameter (units) [Reference range = xx.x to xx.x ]>

| Planned<br>Relative Time | Category | Ambrisentan<br>2.5mg<br>(N=XXX) | Ambrisentan<br>5mg<br>(N=XXX) | Ambrisentan<br>7.5mg<br>(N=XXX) | Ambrisentan<br>10mg<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Baseline** | n | XXX | XXX | XXX | XXX | |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Entry Visit* | n | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Month 3 | n | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Month 6 | n | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | | | | | | |
| Any time<br>Post-baseline | n | XXX | XXX | XXX | XXX | XXX |
| | > reference range high | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | < reference range low | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

For 'Any time in AMB114588 (Entry to End of Study)':-

Subjects with both Normal and Low values are counted once under their worst case (Low).

Subjects with both Normal and High values are counted once under their worst case (High).

Subjects with both High and Low values are counted under both categories.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up. Include Systolic BP, Diastolic BP and Heart Rate.

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Protocol: AMB114588 Population: Safety


Table 3.34: Summary of Physical Examination by Visit

| Planned Relative Time: Entry Visit* | Ambrisentan<br>2.5mg | Ambrisentan<br>5mg | Ambrisentan<br>7.5mg | Ambrisentan<br>10mg | Total<br>(N=XXX) |
|---|---|---|---|---|---|
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| Liver Size | | | | | |
| Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Jugular Venous Pressure | | | | | |
| Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Ascites | | | | | |
| Absent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Present | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Peripheral Oedema | | | | | |
| Absent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Present | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Saturated Oxygen (units) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: \* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588 Population: Safety


Table 3.34: Summary of Physical Examination by Visit

| Planned Relative Time: Month 6 | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|
| | 2.5mg | 5mg | 7.5mg | 10mg | (N=XXX) |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| Liver Size | | | | | |
| N | XX | XX | XX | XX | XX |
| Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal: Improved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal:Unchanged | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal:Worsened | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Jugular Venous Pressure | | | | | |
| N | XX | XX | XX | XX | XX |
| Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal: Improved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal: Unchanged | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal:Worsened | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Ascites | | | | | |
| n | XX | XX | XX | XX | XX |
| Absent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Present: Improved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Present:Unchanged | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Present:Worsened | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Peripheral Oedema | | | | | |
| n | XX | XX | XX | XX | XX |
| Absent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Present: Improved | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal:Worsened | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Abnormal: Unchanged | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588 Population: Safety


Table 3.34: Summary of Physical Examination by Visit

| Planned Relative Time: Month 6 | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|
| | 2.5mg | 5mg | 7.5mg | 10mg | (N=XXX) |
| | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| Saturated Oxygen (units) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: \* Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Safety


Table 3.35: Summary of 12-lead ECG

| Planned<br>Relative Time | Category | Ambrisentan<br>2.5mg | Ambrisentan<br>5mg | Ambrisentan 7.5mg | Ambrisentan<br>10mg | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | |
| Baseline** | n | XXX | XXX | XXX | XXX | XXX |
| baseline | Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | | | | |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| ntry Visít* | n | XXX | XXX | XXX | XXX | XXX |
| - / | Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | , | , , | , , | , | , , | , , |
| onth 6 | n | XXX | XXX | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| onth 12 | n | XXX | XXX | XXX | XXX | XXX |
| Officia 12 | Normal | XX (%) | XXX (%) | XX (%) | XXX (%) | XXX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | ADMOTMAT, CITHICATTY SIGNIFICANC | ΛΛ (δ) | ΛΛ (δ) | AA (6) | ΛΛ (δ) | ΛΛ (δ) |
| tc | | | | | | |
| ny time post-study entry | n | XXX | XXX | XXX | XXX | XXX |
| | Normal | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, not clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | Abnormal, clinically significant | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

For 'Any time in AMB114588 (Entry to End of Study)' if a subject had more than one ECG result, the worst case will be chosen for a conservative approach.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Protocol: AMB114588 Population: Safety


Table 3.36: Summary of Endocrinology assessments - Female

## Overall

| Planned Relative Time | Ambrisentan<br>2.5mg | Ambrisentan<br>5mg | Ambrisentan<br>7.5mg | Ambrisentan<br>10mg | Total |
|---|---|---|---|---|---|
| Baseline** | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Female breast development | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Pre-adolescent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Breast bud stage | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Female pubic hair development | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Pre-adolescent | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Sparse growth | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| Etc | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

 $^{\star}$  Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at baseline: Stage 1 breast development, Post-pubertal at baseline: Stage ≥ 2 breast development.

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present for Baseline, Entry Visit, all available visits, End of Study and Follow Up. Present Overall and by Pubertal Status (Pre-pubertal, Post Pubertal).

Protocol: AMB114588 Population: Safety


Table 3.37: Summary of Endocrinology assessments - Male Overall

| Planned Relative Time | Ambrisentan<br>2.5mg | Ambrisentan<br>5mg | Ambrisentan<br>7.5mg | Ambrisentan<br>10mg | Total |
|---|---|---|---|---|---|
| Baseline** | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Diabt Mastisulas saluma | | | | | |
| Right Testicular volume (units) | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |
| Left Testicular volume | | | | | |
| (units) | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present for Baseline, Entry Visit, all available visits, End of Study and Follow Up. Present Overall and by Pubertal Status (Pre-pubertal, Post Pubertal).

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at baseline: testicular volume < 4 ml, Post-pubertal at baseline: testicular volume ≥ 4 ml

Protocol: AMB114588 Population: Safety


Table 3.37: Summary of Endocrinology assessments - Male Overall

| Planned Relative Time | Ambrisentan<br>2.5mg<br>(N=XXX) | | Ambrisentan<br>5mg<br>(N=XXX) | | Ambrisentan<br>7.5mg<br>(N=XXX) | | | Ambrisentan<br>10mg | | al |
|---|---|---|---|---|---|---|---|---|---|---|
| Baseline** | | | | | | | (N=XXX) | | (N=XXX) | |
| Male genital development | | | | | | | | | | |
| N | XXX | | XXX | | XXX | | XXX | | XXX | |
| Pre-adolescent | XX ( | 응) | XX | (%) | XX | (%) | XX | (%) | XX | (%) |
| Etc | XX ( | 응) | XX | (응) | XX | (응) | XX | (%) | XX | (%) |
| Male pubic hair development | | | | | | | | | | |
| N | XXX | | XXX | | XXX | | XXX | | XXX | |
| Pre-adolescent | XX ( | 응) | XX | (응) | XX | (응) | XX | (%) | XX | (%) |
| Sparse growth | XX ( | 응) | XX | (%) | XX | (%) | XX | (%) | XX | (%) |
| Etc. | XX ( | 응) | XX | (응) | XX | (응) | XX | (%) | XX | (응) |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at baseline: testicular volume < 4 ml, Post-pubertal at baseline: testicular volume ≥ 4 ml

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present for Baseline, Entry Visit, all available visits, End of Study and Follow Up. Present Overall and by Pubertal Status (Pre-pubertal, Post Pubertal).

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Protocol: AMB114588


Population: Safety

Table 3.38: Summary of Pubertal Development Shifts from Baseline - Female Overall

Female Breast Development

| | Planned<br>Relative | Code | Baseline** Code | | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Time | | 1 | 2 | 3 | 4 | 5 |
| Ambrisentan 2.5mg (N=XXX) | Entry<br>Visit* | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/<br>Not Recorded | XX | XX | XX | XX | XX |
| | Etc | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/<br>Not Recorded | XX | XX | XX | XX | XX |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at Baseline: Stage 1 breast development, Post-pubertal at Baseline: Stage ≥ 2 breast development.

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present for Female Breast Development and Female Pubic Hair Development, for each treatment group, overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at all available visits. Put coding below on first page on listing:-

Female Breast Development:-

1=Pre-adolescent; elevation of papilla only, 2=etc...

Female Pubic Hair Development:-

1=Pre-adolescent; vellus over pubes not developed over anterior abdominal wall, 2=etc...

Protocol: AMB114588 Population: Safety


Table 3.39: Summary of Pubertal Development Shifts from Baseline - Male Overall

Male Genital Development

| | Planned<br>Relative | Code | Baseline** Code | | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Time | | 1 | 2 | 3 | 4 | 5 |
| Ambrisentan 2.5mg N=XXX) | Entry<br>Visit* | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/<br>Not Recorded | XX | XX | XX | XX | XX |
| | Etc | 1 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 2 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 3 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 4 | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | 5 | XX (%) | XX (%) | XX (%) | XX (%) | XX |
| | | Unknown/<br>Not Recorded | XX | XX | XX | XX | XX |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at Baseline: testicular volume < 4 ml, Post-pubertal at Baseline: testicular volume ≥ 4 ml

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present for Male Genital Development and Male Pubic Hair Development, for each treatment group, overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at all available visits. Put coding below on first page on listing:-

Male Genital Development:-

1=Pre-adolescent; testes, scrotum and penis same size and proportion, 2=etc...

Male Pubic Hair Development:-

1=Pre-adolescent; velus over pubes no further developed than over abdominal wall, 2=etc...
Protocol: AMB114588 Population: Safety


Table 3.40: Summary of Testicular Volume Change from Baseline - Male Overall

| Planned Relative Time | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| | | 2.5mg | 5mg | 7.5mg | 10mg | |
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Entry Visit* | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Etc | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | ~<br>Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Etc | | | | | | |

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at Baseline: testicular volume < 4 ml, Post-pubertal at Baseline: testicular volume ≥ 4 ml

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at all available visits.

Protocol: AMB114588 Population: Safety


Table 3.41: Summary of Change from Baseline in Plasma Endocrine Parameters - Female Overall

Central Laboratory

Parameter: <Parameter (units)>

| Planned Relative Time | | Ambrisentan | Ambrisentan | Ambrisentan | Ambrisentan | Total |
|---|---|---|---|---|---|---|
| | | 2.5mg | 5mg | 7.5mg | 10mg | |
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| Entry Visit* | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Etc | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Etc | | | | | | |

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at Baseline: Stage 1 breast development, Post-pubertal at Baseline: Stage ≥ 2 breast development.

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit. USER ID: Directory/Program.sas Date Time

Programming notes: Present overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at available visits, for Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B. Change from baseline presented only for the subset of subjects who have QUEST Central labs throughout.

Protocol: AMB114588 Population: Safety


Table 3.42: Summary of Change from Baseline in Plasma Endocrine Parameters - Male Overall

Central Laboratory

Parameter: <Parameter (units)>

| Planned Relative Time | | Ambrisentan<br>2.5mg | Ambrisentan<br>5mg | Ambrisentan<br>7.5mg | Ambrisentan<br>10mg | Total |
|---|---|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) | (N=XXX) |
| | | ***** | ***** | ***** | ***** | |
| Entry Visit* | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Etc | N | XXX | XXX | XXX | XXX | XXX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min. | XX | XX | XX | XX | XX |
| | Max. | XX | XX | XX | XX | XX |
| Etc | | | | **** | | |

Note: \* Entry Visit is at entry to AMB114588.

Baseline is the last value recorded prior to start of study treatment from AMB112529.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Pre-pubertal at Baseline: testicular volume < 4 ml, Post-pubertal at Baseline: testicular volume ≥ 4 ml

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Programming notes: Present overall and by Pubertal Status (Pre-pubertal, Post Pubertal), at available visits, for Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B. Change from baseline presented only for the subset of subjects who have QUEST Central labs throughout.


Protocol: AMB114588

Population: Intent-to-Treat

Table 3.43

Summary of Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to tolerability issues (days)

| | | Ambrisentan Dose Group | | | |
|---|---|---|---|---|---|
| | 2.5mg<br>(N=x) | 5mg<br>(N=xx) | 7.5mg<br>(N=x) | 10mg<br>(N=xx) | Total (N=xx) |
| n | X | × | X | X | х |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | | XX.XX | | xxx.xx4 | XXX.XX |
| Q1 | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x |
| Median | xxx.x | XXX.X | XXX.X | XXXX.X | XXX.X |
| <b>Q</b> 3 | xxx.x | XXX.X | XXX.X | XXXX.X | XXX.X |
| Min. | XXX | XXX | XXX | XXX | XXX |
| Max. | XXX | XXX | XXX | XXXX | XXXX |

Protocol: AMB114588 Page 1 of 36

Table 3.44 Summary of Treatment-Emergent Adverse Events by PAH Therapy

| / | | | | Treatme | ent <i>F</i> | N=10 | 0) | | | Tr | eatment | В (1 | N=100) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | None<br>N=x | | Any<br>N=x | | PDE5<br>Only<br>N=x | 7 | Prost. Only N=x | Both<br>N=x | None<br>N=x | Any<br>N=x | | PDE<br>Onl;<br>N=x | У | Prost. Only N=x | Both<br>N=x |
| ANY EVENT Infections and infestations | X | (100%) | X | (100응) | x | (100%) | 0 | 0 | x (57%) | X | (100%) | х | (100%) | 0 | 0 |
| Any event | X | (100%) | Х | (67%) | х | (67%) | 0 | 0 | x (29%) | X | (67%) | X | (67%) | 0 | 0 |
| Upper respiratory tract infection | | (100%) | | (33%) | | (33%) | | 0 | x (14% | | (22%) | | (22%) | 0 | 0 |
| Nasopharyngitis | 0 | | 0 | | 0 | | 0 | 0 | x (14%) | Х | (44%) | X | (44%) | 0 | 0 |
| Pharyngitis | 0 | | X | (33%) | X | (33%) | 0 | 0 | 0 | X | (33%) | Х | (33%) | 0 | 0 |
| Gastroenteritis | 0 | | X | (33%) | X | (33%) | 0 | 0 | 0 | X | (22%) | Х | (22%) | 0 | 0 |
| Influenza | 0 | | 0 | | 0 | | 0 | 0 | 0 | X | (33%) | Х | (33%) | 0 | 0 |
| Pneumonia | 0 | | X | (33%) | 1 | (33%) | 0 | 0 | 0 | X | (11%) | Х | (11%) | 0 | 0 |
| Bronchitis | 0 | | 0 | | 0 | | 0 | 0 | 0 | X | (11%) | X | (11%) | 0 | 0 |
| Gastroenteritis viral | 0 | | 0 | | 0 | | 0 | 0 | 0 | X | (22%) | X | (22%) | 0 | 0 |
| Hordeolum | 0 | | 0 | | 0 | | 0 | 0 | 0 | X | (11%) | X | (11%) | 0 | 0 |
| Otitis externa | 0 | | 0 | | 0 | | 0 | 0 | 0 | X | (22%) | X | (22%) | 0 | 0 |
| Otitis media | 0 | | 1 | (33%) | X | (33%) | 0 | 0 | 0 | 0 | | 0 | | 0 | 0 |
| Otitis media chronic | 0 | | 1 | (33%) | Х | (33%) | 0 | 0 | 0 | 0 | | 0 | | 0 | 0 |
| Pharyngotonsillitis | 0 | | 0 | | 0 | | 0 | 0 | 0 | 0 | | 0 | | 0 | 0 |
| Respiratory tract infection | 0 | | 0 | | 0 | | 0 | 0 | 0 | 0 | | 0 | | 0 | 0 |
| Rhinitis | 0 | | 0 | | 0 | | 0 | 0 | 0 | Х | (11%) | X | (11%) | 0 | 0 |
| Sinusitis | 0 | | 0 | | 0 | | 0 | 0 | 0 | 1 | (11%) | Х | (11%) | 0 | 0 |

Note: Prost.=Prostanoids.

USER ID: Directory/Program.sas Date Time

## Programming Notes: Repeat for

Population: Safety

| 3.45 | Summary of Serious Treatment Emergent Adverse Events by PAH Therapy |
|---|---|
| 3.46 | Summary of Non-Serious Treatment Emergent Adverse Events by PAH Therapy |
| 3.47 | Summary of Common (>=5%) Treatment Emergent Adverse Events by PAH Therapy Footnote: Note: Common adverse events (>=5%) were those experienced by at least 5% of subjects in the total population (N=38) irrespective of dose group and/or PAH therapy |

|-----|--------------|-----------|

Protocol: AMB114588 Page 1 of xx

Table 3.48
Summary of Treatment Emergent Adverse Events by PAH Aetiology

| | Treatment A (N=100) Non- Idiopathic Idiopathic N=xx N=xx | | Treatment B (N= | =100) | Treatment C (N=6) | |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | | | Idiopathic<br>N=xx | Non-<br>Idiopathic<br>N=xx | Idiopathic<br>N=xx | Non-<br>Idiopathic<br>N=xx |
| ANY EVENT | <br>0 | <br>х (хх%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Infections and infestations | | | | | | |
| Any event | 0 | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Upper respiratory tract infection | 0 | x (xx%) | x (xx%) | x (xx%) | x (xx%) | x (xx%) |
| Nasopharyngitis | 0 | 0 | x (xx%) | x (xx%) | x (xx%) | 0 |
| Pharyngitis | 0 | x (xx%) | x (x%) | x (xx%) | 0 | 0 |
| Gastroenteritis | 0 | x (xx%) | 0 | xx (xx%) | 0 | 0 |
| Influenza | 0 | 0 | x (xx%) | x (xx%) | 0 | 0 |
| Bronchitis | 0 | 0 | 0 | 1 (xx%) | x (xx%) | 0 |
| Gastroenteritis viral | 0 | 0 | x (x%) | 1 (xx%) | 0 | 0 |
| Hordeolum | 0 | 0 | 0 | 1 (xx%) | 1 (xx%) | 0 |
| Otitis externa | 0 | 0 | 0 | 2 (xx%) | 0 | 0 |
| Otitis media | 0 | x (xx%) | 0 | 0 | 0 | 0 |

Note: Idiopathic group refers to those with an idiopathic aetiology of PAH at baseline in study AMB112529 and non-idiopathic refers to those classified as having an aetiology of familial, persistent PAH despite surgical repair, or secondary to connective tissue disease.

USER ID: Directory/Program.sas Date Time

## Programming Notes:

Population: Safety

Repeat for

| 3.49 | Summary of Serious Treatment Emergent Adverse Events by PAH Aetiology |
|---|---|
| 3.50 | Summary of non-Serious Treatment Emergent Adverse Events by PAH Aetiology |
| 3.51 | Summary of Common (>=5%)Treatment Emergent Adverse Events by PAH Aetiology Footnote: Note: Common adverse events (>=5%) were those experienced by at least 5% of subjects in the total population (N=38) irrespective of dose group and/or PAH Aetiology. |

| RAP |
|-----|
|-----|

Protocol: AMB114588 Population: Safety

Table 3.52 Summary of Cardiopulmonary Hemodynamics

| Parameter | Treatment | Planned<br>Relative Time | n | Mean | SD | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| <parameter (units)=""></parameter> | Ambrisentan<br>2.5mg | Baseline** | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | (N=XXX) | Entry Visit | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 3 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 6 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 9 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Month 12 | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | | Etc | XXX | XX.X | XX.XX | XX.X | XX.X | XX.X | XX | XX |
| | Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| | Ambrisentan<br>5mg<br>(N=XXX) | Etc | | | | | | | | |
| | Ambrisentan<br>5mg | Etc | | | | | | | | |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

USER ID: Directory/Program.sas Date Time

Programming notes: Present available visits, End of Study and Follow-Up. Include all the available parameters.

<sup>\*</sup> Entry Visit is at entry to AMB114588.

Q1 = 1st quartile, Q3 = 3rd quartile.

Subjects are considered as belonging to the treatment group according to the highest dose received.

Protocol: AMB114588

Population: Intent-to-Treat

Listing 1.1: Listing of Reasons for Study Withdrawal


Treatment: Ambrisentan 2,5mg

| Centre ID/ | Date of | Study | Reason for |
|------------|------------|-------|--------------|
| Subject ID | Withdrawal | Day | Withdrawal |
| XXXXXX/ | DDMMMYYYY | XX | XXXXXXXXXXXX |
| XXXXXX | | | |
| XXXXXX/ | DDMMMYYYY | XX | XXXXXXXXXXXX |
| XXXXXX | | | |
| XXXXXX/ | DDMMMYYYY | XX | XXXXXXXXXXXX |
| XXXXXX | | | |
| Etc | | | |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.2: Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Type | Criterion |
|---|---|---|
| XXXXXX/<br>XXXXXX | Inclusion | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | Exclusion | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Listing 1.3: Listing of Demographic Characteristics

Treatment: Ambrisentan 2,5mg

| / | Centre ID/<br>Subject ID | Partial<br>Date of Birth | Age (years)* | Sex | Child Bearing<br>Potential | Has Child<br>Bearing<br>Potential<br>Changed? | Date of Child<br>Bearing<br>Potential<br>Change | Ethnicity |
|---|---|---|---|---|---|---|---|---|
| | XXXXXX/<br>XXXXXX | YYYY | XX | Female | Pre-menarcheal | Yes | DDMMMYYYY ^ | Hispanic/Latino |

Etc..

Note: \* Age at start of study treatment in AMB112529

- ^ Date of first menses
- # Date of final menses
- ~ Date became sterile

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.4: Listing of Race

Treatment: Ambrisentan 2,5mg

Centre ID/ Subject ID Race

XXXXXX/ XXXXXX Asian - East Asian Heritage

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time


Population: Intent-to-treat

Listing 1.5: Listing of Disease History

Treatment: Ambrisentan 2,5mg

| Centre ID /<br>Subject ID | Diagnosis | Sub category | Date of<br>Diagnosis | Duration<br>of PAH<br>(yrs) | Baseline<br>WHO FC |
|---|---|---|---|---|---|
| xxxxxx / | Idiopathic PAH | | DDMMMYYYY | Х.Х | I |
| xxxxxx /<br>xxxxxx | Persistent PAH despite surgical repair | Atrio-ventricular septal defects | DDMMMYYYY | Х.Х | II |
| Etc | | | | | |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID. Produce listing for data collected in AMB112529 for the subset of subjects who entered AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.6: Listing of Medical Conditions

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/ | Classification | Preferred Term | Condition | Status |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX | Hepatobiliary disorders | xxxxxxxxxxxx | HEPATITIS A | Current |
| | | Psychiatric disorders | xxxxxxxxxxxx | PARANOIA COMBINED WITH MANIA. | Past |
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX | Eye disorders | XXXXXXXXXXXXXXX | ASTIGMATISM | Current |
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX | Metabolism and nutrition disorders | XXXXXXXXXX | RICKETS | Current |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID. Produce listing for data collected in AMB112529 for the subset of subjects who entered AMB114588.

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.7: Listing of Medications

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | | Total<br>Daily | | | |
|---|---|---|---|---|---|
| Subject ID | ATC Level 1/<br>Ingredient/<br>Verbatim Text | Daily<br>Dose/<br>Units/<br>Freq/<br>Route | Date<br>Started/<br>Study Day | Date<br>Stopped/<br>Study Day | Reason<br>For<br>Medication |
| XXXXXX/<br>XXXXXX | <pre>Endocrine &amp; metabolic/ Fluticasone propionate/ FLIXOTIDE #</pre> | 2/<br>MG/<br>2XD/<br>IH | 27SEP1999/<br>15 | 020CT1999 | xxxxxxxxx |
| | <pre>Endocrine &amp; metabolic/ Fluticasone propionate/ FLIXOTIDE #</pre> | 4/<br>MG/<br>2XD/<br>IH | 03OCT1999/<br>21 | Ongoing | |
| | E+ c | | | | |

Etc..

Etc..

Note: \* Prior, # Concomitant, \$ Post-treatment.

PAH Therapies are not included within this listing, for PAH Therapy please see Listing 1.7 Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Listing 1.8: Listing of PAH Therapy

Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Drug Class/<br>ATC Level 1/<br>Ingredient/<br>Verbatim Text/ | Total<br>Daily<br>Dose/<br>Units | Date<br>Started/<br>Study Day | Date<br>Stopped/<br>Study Day | Reason the medication started? |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X/<br>XX | DDMMMYYYY/<br>XX | DDMMMYYYY | xxxxxxxxxxxx |
| XXXXXX/<br>XXXXXX | XXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXX | X/<br>XX | DDMMMYYYY/<br>XX | Ongoing | XXXXXXXXXXXX |
| | Etc | | | | |

Etc..

Note: \* Prior, # Concomitant, \$ Post-treatment.

@ Ongoing background PAH therapy at baseline

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|

Population: Intent-to-Treat


Listing 1.9: Relationship between ATC Level 1, Ingredient and Verbatim Text

| ATC Level 1 | Ingredient | Verbatim Text |
|---|---|---|
| Endocrine & metabolic | Fluticasone Propionate<br>Prednisolone | FLIXOTIDE<br>PREDNISOLONE |
| Drugs acting via the nervous system | Paracetamol | PANADOL<br>CHILDREN'S PANADOL 1-5YERS |
| Etc | | |

USER ID: Directory/Program.sas Date Time

Programming notes: Sort by ATC level 1treatment group, Ingredient.

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.10: Listing of Compliance Data

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | % of compliant visits | Visit | Visit Date/<br>Study Day | Compliance since the last visit |
|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | 100 | XXXXXXXX | DDMMMYYYY/<br>XX | |
| | | XXXXXXXX | DDMMMYYYY/<br>XX | >=80% and <=120% |

Etc..

Note: Compliant visits are those at which subjects are >=80% and <=120% compliant.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.11: Listing of initial, highest and final dose of ambrisentan

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Initial dose mg/kg | Highest dose mg/kg | Final dose mg/kg |
|---|---|---|---|
| XXXXXX/<br>XXXXXX | х.х | х.х | x.x |
| XXXXXX/<br>XXXXXX | х.х | X.X | х.х |
| | Etc | | |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 1.12: Listing of Protocol Deviation

Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Important<br>Protocol<br>Deviations | Protocol Deviation Category | Protocol Deviation<br>Description | Protocol<br>Deviation Date/<br>Study Day | Visit<br>Phase | Action<br>taken | Escalated for Medical Oversight? |
|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | Y | Biological specimen sample procedures | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>XX | XXXXXXXX | XXXXXXXXX<br>XXXXXXXX<br>XXXXX | |
| XXXXXX/<br>XXXXXX | N | Other:<br>XXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXXXX<br>XXXXXXXX<br>XXXXX | |
| | | Etc | | | | | |

Etc..

Note: \* Important Deviation

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 2.1: Listing of Time to Death (All cause)

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Death Date/<br>Study Day | Details |
|--------------------------|--------------------------|---------|
| XXXXXX/ | DDMMMYYYY/ | |
| XXXXXX | XX<br>DDMMMYYYY/ | |
| | XX | |
| Etc | | |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Listing 2.2: Listing of 6 Minute Walking Distance Data

Treatment: Ambrisentan 2,5mg

| Centre | | | Di | stance Walke | ed (m) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| ID/<br>Subject<br>ID | Visit | Visit Date/<br>Time/<br>Study Day | Actual | Change<br>from<br>Baseline | Percentage<br>Change<br>from<br>Baseline | Did subject walk less than 6 minutes?/ Reason for stopping prematurely | Duration<br>walked<br>(seconds) | Did subject<br>use<br>supplemental<br>oxygen | Oxygen<br>flow<br>rate<br>(L/min) |
| XXXXXX/<br>XXXXXX | Baseline ** | DDMMMYYYY/<br>HH:MM/<br>XX | XXX | | | Y/<br>XXXXXXXXXXXX | XXX | У | XXXX |
| | Entry Visit * | DDMMMYYYY/<br>HH:MM/<br>XX | XXX | XXX | XXX | Y/<br>XXXXXXXXXXXX | XXX | Y | XXXX |
| | XXXXXXX | DDMMMYYYY/<br>HH:MM/<br>XX | XXX | XXX | XXX | N | | N | |
| | XXXXXX | DDMMMYYYY/<br>HH:MM/<br>XX | XXX | XXX | XXX | N | | N | |
| | Etc | | | | | | | | |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Listing 2.3: Listing of Clinical Worsening of PAH

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Event Date/<br>Study Day | Clinical worsening criteria |
|---|---|---|
| XXXXXX/ | DDMMMYYYY/ | Hospitalisation for worsening of PAH |
| XXXXXX | XX<br>DDMMMYYYY/<br>XX | PAH related deterioration: Clinical signs or symptoms of right sided heart failure |
| Etc | | |

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|

Population: Intent-to-Treat


Listing 2.6: Listing of WHO Functional Class Data

Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Visit | Visit<br>Date/<br>Study Day | WHO pulmonary hypertension functional classification | Actual \$ | Change<br>from<br>Baseline | Change<br>Categorisatio<br>n |
|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | Baseline ** | DDMMMYYYY/<br>XX | Class II | 2 | | |
| ΛΛΛΛΛ | Entry Visit * | DDMMMYYYY/<br>XX | Class II | 2 | 0 | NC |
| | XXXXXXX | DDMMMYYYY/<br>XX | Class IV | 4 | 2 | Det |
| | XXXXXX | DDMMMYYYY/<br>XX | Class I | 1 | -1 | Imp |
| | Etc | | | | | |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

There are 4 grades for WHO FC based on severity of symptoms (\$\frac{1}{2}\$\$ \$ Grades mapped to numeric scale 1-4 (i.e. Class IV = 4).

Change categorisation (based on -2, -1, 0, +1, +2);

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Listing 2.7: Listing of Plasma NT-Pro BNP Concentration (ng/L)

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Visit | Visit<br>Date/<br>Study Day | Value | Change from Baseline | | |
|---|---|---|---|---|---|---|
| | | | Raw | Log | Raw | Log\$ |
| XXXXXX/<br>XXXXXX | Baseline ** | DDMMMYYYY/<br>XX | XXX.X | X.XX | | |
| | Entry Visit * | DDMMMYYYY/<br>XX | XXX.X | X.XX | XXX.X | X.XX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX.X | X.XX | XXX.X | X.XX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXX.X | X.XX | XXX.X | X.XX |
| | Etc | | | | | |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

- \* Entry Visit is at entry to AMB114588.
- \$ Log (change from baseline) = Log (Visit) Log (Baseline).
- Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 2.8: Listing of Exploratory Echocardiogram

Treatment: Ambrisentan 2,5mg

| Centre<br>ID/<br>Subject<br>ID | Visit | Visit<br>Date/<br>Study Day | Pericardial<br>effusion/<br>Change from<br>Baseline | Mean right atrial pressure (mmHg)/Change from Baseline | Tricuspid annular plane systolic excursion (cm)/ Change from Baseline | Systolic<br>Eccentricity<br>Index/<br>Change from<br>Baseline | Diastolic<br>Eccentricity<br>Index/<br>Change from<br>Baseline | Tricuspid<br>regurgitant<br>jet (m/s)/<br>Change from<br>Baseline | Right Ventricular Pressure (mmHg)/ Change from Baseline |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | Baseline<br>** | DDMMMYYYY/<br>XX | Absent | XXX | XXX | XXX | XXX | XXX | XXX |
| 2171217121 | Entry | DDMMMYYYY/ | Trace/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | Visit * | XX | Worsened | XXX | XXX | XXX | XXX | XXX | XXX |
| | XXXXXXX | DDMMMYYYY/ | Small/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | XX | Worsened | XXX | XXX | XXX | XXX | XXX | XXX |
| | XXXXXXX | DDMMMYYYY/ | Trace/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | | XX | Worsened | XXX | XXX | XXX | XXX | XXX | XXX |
| | Etc | | | | | | | | |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 2.9: Listing of Cardiopulmonary Hemodynamics

Treatment: Ambrisentan 2,5mg

| Centre ID/ | | | | | |
|---|---|---|---|---|---|
| Subject ID | Right Heart Catheterization Date / Time/ Study Day | Heart<br>Rate(bpm)/<br>Change from<br>Baseline | Mean Pulmonary<br>Arterial<br>Pressure (mmHg)/<br>Change from<br>Baseline | Mean Right Atrial Pressure (mmHg)/ Change from Baseline | Pulmonary<br>Capillary Wedge<br>Pressure (mmHg)/<br>Change from<br>Baseline |
| VVVVVVVV / | DDMMMM37373737 / | 77777 | 77777 | 7777 | 7777 |
| XXXXXX/<br>XXXXXX | DDMMMYYYY/<br>HH:MM/<br>XX | XXX | XXX | XXX | XXX |
| | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | HH:MM/<br>XX | XXX | XXX | XXX | XXX |
| | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | HH:MM/<br>XX | XXX | XXX | XXX | XXX |
| | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | HH:MM/<br>XX | XXX | XXX | XXX | XXX |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 2.9: Listing of Cardiopulmonary Hemodynamics

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Right Heart<br>Catheterization<br>Date /<br>Time/<br>Study Day | Method used to<br>Calculate<br>Cardiac Output/<br>Oxygen<br>Consumption | Cardiac Output<br>(Litres/minute)/<br>Change from<br>Baseline | Cardiac index (L/min/meters/ square)/Change from Baseline | Pulmonary Vascular<br>Resistance<br>(mmHg/L/min)/<br>Change from<br>Baseline |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | DDMMMYYYY/<br>HH:MM/<br>XX | xxxxxxxxxxx/<br>xxxxxxxxxxxx | XXX | xxx | xxx |
| | DDMMMYYYY/<br>HH:MM/<br>XX | XXXXXXXXXXX/<br>XXXXXXXXXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| | DDMMMYYYY/<br>HH:MM/<br>XX | XXXXXXXXXXX/<br>XXXXXXXXXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |
| | DDMMMYYYY/<br>HH:MM/<br>XX | XXXXXXXXXXX/<br>XXXXXXXXXXX | XXX/<br>XXX | XXX/<br>XXX | XXX/<br>XXX |

Etc..

Note: Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 2.9: Listing of Cardiopulmonary Hemodynamics

Treatment: Ambrisentan 2,5mg

| Centre ID/ | | | Arterial | | |
|---|---|---|---|---|---|
| Subject ID | Right Heart | Left Ventricle | Oxygen | Venous | |
| | Catheterization | End Diastolic | Saturation | Oxygen | Mean Arterial |
| | Date / | Pressure (mmHg)/ | Percentage/ | Saturation/ | Pressure (mmHg)/ |
| | Time/ | Change from | Change from | Change from | Change from |
| | Study Day | Baseline | Baseline | Baseline | Baseline |
| XXXXXX/ | DDMMMYYYY **/ | XXX | XXX | XXX | XXX |
| XXXXXX | HH:MM/ | 11111 | 212121 | 212121 | |
| | XX | | | | |
| | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | HH:MM/ | XXX | XXX | XXX | XXX |
| | XX | | | | |
| | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | HH:MM/ | XXX | XXX | XXX | XXX |
| | XX | | | | |
| | DDMMMYYYY/ | XXX/ | XXX/ | XXX/ | XXX/ |
| | HH:MM/ | XXX | XXX | XXX | XXX |
| | XX | | | | |

Etc..

Note: \*\* Baseline - the last value recorded prior to start of study treatment from AMB112529.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Intent-to-Treat


Listing 2.10: Listing of School Days

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Visit Date<br>/<br>Study Day | School Days<br>Scheduled/<br>Change from<br>Baseline | School Days<br>missed/<br>Change from<br>Baseline | School Days<br>missed due<br>to PAH/<br>Change from<br>Baseline | Proportion of days missed (%)/<br>Change from Baseline | Proportion of<br>days missed due<br>to PAH (%)/<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>Male/<br>XXXXXX | Baseline ** | DDMMMYYYY/<br>XX | XX | XX | XX | XX | XX |
| | | Entry | DDMMMYYYY/ | XX/ | XX/ | XX/ | XX/ | XX/ |
| | | Visit * | XX | XX | XX | XX | XX | XX |
| | | XXXXXXX | DDMMMYYYY/ | XX/ | XX/ | XX/ | XX/ | XX/ |
| | | | XX | XX | XX | XX | XX | XX |
| | | XXXXXXX | DDMMMYYYY/ | XX/ | XX/ | XX/ | XX/ | XX/ |
| | | | XX | XX | XX | XX | XX | XX |
| | | | XX | XX | XX | XX | XX | 2 |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

Etc..

\* Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Population: Intent-to-Treat


Listing 2.11: Listing of Subject Global Assessment (SF10 Health Survey for Children)

Treatment: Ambrisentan 2,5mg

Centre ID/ Subject ID

| | Visit | Visit Date /<br>Study Day | 1.Childs General<br>Health | 2a.Limited Riding and Skating | 2b.Limited<br>Bending | 3.Physical<br>Problems Limit<br>Schoolwork | 4.Emotional Problems Limit Schoolwork | 5.Bodily pain |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | Baseline<br>** | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | xxxxxxx |
| | Entry<br>Visit * | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |
| | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

The Physical Summary Score (aggregate of item responses 1, 2a, 2b, 3 and 5) and Psychosocial Summary Score (aggregate of item responses 4, 6, 7, 8 and 9) were calculated by QualityMetrics Health Outcomes software. Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Etc..

Population: Intent-to-Treat


Listing 2.11: Listing of Subject Global Assessment (SF10 Health Survey for Children)

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Visit | Visit Date<br>/<br>Study Day | 6.Satisfied with friendships | 7.Satisfied with life overall | 8.Time bothered or upset | 9.General<br>behaviour | Physical<br>Health<br>Summary/<br>Change<br>from<br>Baseline | Psychosocial<br>Summary/<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/ | Baseline ** | DDMMMYYYY/ | XXXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XX | XX |
| XXXXXX | | XX | | | | | | |
| | Entry Visit | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XX/ | XX/ |
| | * | XX | | | | | XX | XX |
| | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XX/ | XX/ |
| | | XX | | | | | XX | XX |
| | XXXXXXX | DDMMMYYYY/ | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XX/ | XX/ |
| | | XX | | | | | XX | XX |
| | Etc | | | | | | | |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

The Physical Summary Score (aggregate of item responses 1, 2a, 2b, 3 and 5) and Psychosocial Summary Score (aggregate of item responses 4, 6, 7, 8 and 9) were calculated by QualityMetrics Health Outcomes software.

Subjects are considered as belonging to their treatment group at the start of study AMB114588.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Safety

Listing 3.1: Listing of Exposure Investigational Product

Treatment: Ambrisentan 2,5mg

| Subject<br>ID | IP<br>Start<br>Date | IP<br>Stop<br>Date | Duration<br>(Months) | Start Date<br>of Dose/<br>Study Day | End Date<br>of Dose /<br>Study Day | Dose | Dose<br>Unit | Primary reason for change |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | DDMMMYYYY | DDMMMYYYY | XXX | DDMMMYYYY/<br>XX | DDMMMYYYY/<br>XX | Χ^ | XX | |
| | | | | DDMMMYYYY/<br>XX | DDMMMYYYY/<br>XX | Χ^ | XX | XXXXXXXXXX |
| | | | | DDMMMYYYY/<br>XX | DDMMMYYYY/<br>XX | Χv | XX | XXXXXXXXXX |

Etc..

Note: ^ Up titration, v Down titration, # Restart of investigational product.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group, subject and time-point.


Population: Safety

Listing 3.2: Listing of All Adverse Events

| Treatment: Ambriser | ntan 2 5mg | | | 110cmg 3.2. 110 | cing of hir haven | DC DVCIICD | | |
|---|---|---|---|---|---|---|---|---|
| Treatment. Ambitser | Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/<br>Weight<br>(kg) | Preferred Term/<br>Verbatim Text | Outcome/<br>Onset Date/<br>Resolution Date/<br>Frequency | Time Since<br>First Dose/<br>Last Dose/<br>Duration (days) | Maximum<br>Intensity/<br>Serious/<br>Withdrawal | Action<br>Taken/<br>Relation to<br>Study Drug | Further Details if<br>Serious Event |
| | XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/<br>XXXXXX/<br>XX | XXXXXXXXXXX/<br>XXXXXXXXXXX * | XXXXXXXX/ DDMMMYYYY/ DDMMMYYYY/ XXXXXXXXX | XX/<br>XX/<br>XX | XXXX/<br>XXX/<br>XXX | XXXXXXX/<br>XX | e.g. Results in death, Results in disability/ Incapacity, Congential anomaly/ birth defect, Possible drug induced liver injury, Life threatening, Requires prolonged hospitalisation, Caused by activity related to study, Etc |
| | | | XXXXXXXXXX/<br>XXXXXXXXXX # | XXXXXXXX/ DDMMMYYYY/ DDMMMYYYY/ XXXXXXXXX | XX/<br>XX/<br>XX | XXXX/<br>XXX/<br>XXX | XXXXXXX/<br>XX | |
| | XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/<br>XXXXXX/<br>XX | XXXXXXXXXXX/<br>XXXXXXXXXXX \$ | XXXXXXXX/ DDMMMYYYY/ DDMMMYYYY/ XXXXXXXXX | XX/<br>XX/<br>XX | XXXX/<br>XXX/<br>XXX | XXXXXXXX/<br>XX | |

Etc..

Note: \* Prior, # Treatment-emergent, \$ Post-treatment, ~ AE started pre extension study.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|
|-----|--------------|-----------|

Protocol: AMB114588 Population: Safety


Listing 3.3: Listing of Relationship between Adverse Event System Organ Class, Preferred Term and Verbatim Text

| System Order Class | Preferred Term | Verbatim Text |
|---|---|---|
| Blood and lymphatic system<br>disorder | Lymphadenopathy | Enlarged lymph node |
| Cardiac disorder | Palpitations<br>Tachycardia nos | Heart palpitation<br>Tachycardia |
| Etc | | |

USER ID: Directory/Program.sas Date Time

Programming notes: Continue for all combinations. Sort in order of SOC, PT, and verbatim text.

| F | RAP | CONFIDENTIAL | AMB114588 | l |
|---|-----|--------------|-----------|---|
|---|-----|--------------|-----------|---|

Protocol: AMB114588


Population: Safety

Listing 3.4: Listing of Subject Numbers for Specified Adverse Events

Treatment: Ambrisentan 2,5mg

| System Organ Class | No. with | Centre ID/Subject ID |
|---|---|---|
| Preferred term | Event | |
| Gastrointestinal disorders | | |
| Dyspepsia | 9 | XXXXXX/XXXXXX, |
| Nausea<br>Etc | 1 | XXXXXX/XXXXXX |

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group. Sort by treatment group, SOC, PT.


Population: Safety

Listing 3.8: Listing of Haematology

Central / Local Laboratory
Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race/ | | Planned | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseline | | Relative | | Study | Converte | Flag \$ | | |
| | Weight(kg) | Lab test (units) | Time | Date | Day | Value | Normal Range | NR C | CC BL |
| XXXXXX/<br>XXXXXX | XX/ | <parameter (units)=""></parameter> | Baseline ** | DDMMMYYYY | XX | XXX | XXX - XXX | | |
| | XXXXXX/ | | Entry Visit* | DDMMMYYYY | XX | XXX | XXX - XXX | | |
| | XXXXXX/ | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | H F | Н Н |
| | XX | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | Н | Н |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | | |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | | |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | | |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | L I | ı L |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | | |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | L | |

<Parameter (units)> Etc..

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

\$ NR for Normal Range flag, CC for Clinical Concern flag; BL for Change from Baseline

H=Above range, L=Below range

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time
Protocol: AMB114588 Population: Safety


Listing 3.9 Listing of Haematology Data for Subjects with Abnormalities of Potential Clinical Concern

Central /Local Laboratory
Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race/ | | Planned | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline | | Relative | | Study | Conver | ted Data | | | Fl | ag S | \$ |
| | Weight(kg) | Lab test (units) | Time | Date | Day | Value | Normal<br>Range | Low<br>Concern | High<br>Concern | _ | сс | |
| XXXXXX/<br>XXXXXX | XX/ | <parameter (units)=""></parameter> | Baseline<br>** | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | XXXXXX/ | | Entry<br>Visit* | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | XXXXXX/ | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | Н | Н | Н |
| | XX | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | Н | | Н |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | XXXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | XXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | XXXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | L | L | L |
| | | | XXXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | | | |
| | | | XXXXXXXXX | DDMMMYYYY | XX | XXX | XXX - XXX | XXX | XXX | L | | |

<Parameter (units)> Etc..

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

\$ NR for Normal Range flag, CC for Clinical Concern flag; BL for Change from Baseline

H=Above range, L=Below range

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

| RAP |
|-----|
|-----|

Protocol: AMB114588

Population: Safety


Listing 3.13: Listing of Liver Event Results and Time of Event Relative to Treatment

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/ | Event Date/<br>Study Day | Days from<br>first dose to<br>start of<br>event | Days from last dose to start of event | Event that reached or exceeded protocol defined criteria |
|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/ | DDMMMYYYY/ | X | X | ALT (alanine aminotransferase) |
| | XXXXXX/<br>XXXXXX/<br>XX | XX | | | |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

| .P | CONFIDENTIAL | AMB114588 |
|----|--------------|-----------|
|----|--------------|-----------|

Population: Safety

Listing 3.14: Listing of patient specific information for liver events

Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/ | Event that reached or exceeded protocol defined criteria | Event Date/<br>Study Day | Days from last dose to start of | | |
|---|---|---|---|---|---|---|
| | | | | event | Assessment | Result |
| XXXXXX/<br>XXXXXX | XX/ | XXXXXXXXXXX | DDMMMYYYY/ | X | Subject become pregnant? | No |
| | XXXXXX/<br>XXXXXX/<br>XX | | XX | | Was a biopsy taken? Any unconventional medications Fasting or significant dietary change Is this event serious? Evaluation interval | Yes No No Yes During the treatment period |
| | | | | | Does the subject consume alcohol? Average number of units of alcohol consumed per week | Yes<br>XX |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

| RAP |
|-----|
|-----|

Protocol: AMB114588 Population: Safety


Listing 3.15: Listing of Medical Conditions for Subjects with Liver Events on Treatment

| Treatment | Centre<br>ID/<br>Subject<br>ID | Age (y)/<br>Sex/<br>Race/ | Classification | Condition | Status |
|---|---|---|---|---|---|
| Ambrisentan<br>2.5mg | XXXXXX/<br>XXXXXX | XX/<br>XXXXXXX/<br>XXXXXX | Hepatobiliary | HEPATITIS A | Current |
| | | | Psychiatric | PARANOIA COMBINED WITH MANIA. | Past |
| | XXXXXX/<br>XXXXXX | XX/<br>XXXXXXX/<br>XXXXXX | Eye | ASTIGMATISM | Current |
| Ambrisentan<br>5mg | XXXXXX/<br>XXXXXX | XX/<br>XXXXXXX/<br>XXXXXX | Metabolism and nutrition | RICKETS | Current |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

|------------------------|
|------------------------|

Protocol: AMB114588

Protocol: AMB114388

Population: Safety

Listing 3.16: Listing of Liver Biopsy Details


Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/ | Event that reached or exceeded protocol defined criteria | Biopsy Date/<br>Study Day | Biopsy<br>Size<br>(mm) | Liver biopsy test | Liver biopsy result |
|---|---|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/ | xxxxxxxxxxx | DDMMMYYYY/ | X | Bile ducts | Other: Bile ducts blocked |
| | XXXXXX/<br>XXXXXX/<br>XX | | XX | | Final diagnosis Description of liver cells/hepatocytes Liver cell/hepatocyte inclusion/vacuole Hepatocyte/liver cell nuclear abnorm Etc | Alcoholic hepatic cirrhosis<br>Normal<br>No inclusions<br>None |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

Population: Safety

Listing 3.17: Listing of Liver Imaging Details

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Age (y)/<br>Sex/<br>Race/ | Event that reached or exceeded protocol defined criteria | Imaging Date/<br>Study Day | Liver<br>imaging | Are images<br>technically | | |
|---|---|---|---|---|---|---|---|
| | | | | method | adequate? | Liver imaging test | Liver imaging result |
| XXXXXX/<br>XXXXXX | XX/ | XXXXXXXXXXX | DDMMMYYYY/ | X | XX | Liver Size | Hypertrophy (or enlarged) |
| AAAAA | XXXXXX/<br>XXXXXX/ | | XX | | | Liver Texture | Normal |
| | ******* | | | | | Liver fatty infiltrate grade | Not applicable - No fatty<br>infiltration |
| | XX | | | | | Ascites present | None present |
| | | | | | | Focal hepatic lesions character | Not applicable - no hepatic lesions |
| | | | | | | Gallstones or gallbladder lesions | None |
| | | | | | | Biliary ductal lesions | None |
| | | | | | | Portal/Hepatic vein abnormalities | None |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Present each treatment group and Centre/Subject ID. Sort by treatment group, Centre ID, Subject ID.

|-----|--------------|-----------|

Population: Safety

Listing 3.18: Listing of Vital Signs

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | Age(y)/ | | Visit | Systolic<br>Blood<br>Pressure<br>(mmHg) /<br>Change | Diastolic<br>Blood<br>Pressure<br>(mmHg)/<br>Change | Heart<br>Rate<br>(bpm)/<br>Change | Height (units)/Change | Weight (units)/ Change | BMI<br>(units)/<br>Change | BSA (units)/Change |
|---|---|---|---|---|---|---|---|---|---|---|
| | Sex/<br>Race | Visit | Date/<br>Study Day | from<br>Baseline | from<br>Baseline | from<br>Baseline | from<br>Baseline | from<br>Baseline | from<br>Baseline | from<br>Baseline |
| | Nace | VISIC | Scuay Day | Daseiille | Daseiille | Daseille | Daseiille | Daseiille | Daseiille | Daseille |
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/ | Baseline ** | DDMMMYYYY/<br>XX | XX | XX | XX | XX | XX | XX | XX |
| | XXXXXX | Entry | DDMMMYYYY/ | XX/ | XX/ | XX/ | XX/ | XX/ | XX/ | XX/ |
| | | Visit * | XX | XX | XX | XX | XX | XX | XX | XX |
| | | XXXXXXX | DDMMMYYYY/ | XX/ | XX/ | XX/ | XX/ | XX/ | XX/ | XX/ |
| | | | XX | XX | XX | XX | XX | XX | XX | XX |

Etc..

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

H=Above clinical concern, L=Below clinical concern,

Change from Baseline HC=Above clinical concern, LC=Below clinical concern

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|

Protocol: AMB114588

Population: Safety

Listing 3.20: Listing of Physical Examination


Treatment: Ambrisentan 2.5mg

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Visit<br>Date/<br>Study Day | Liver<br>Size | Jugular<br>Venous<br>Pressure | Ascites | Peripheral<br>Oedema | Saturated<br>Oxygen<br>(units) |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/ | XX/ | Entry | DDMMMYYYY/ | XXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XX.XXX |
| XXXXXX | XXXXXX/<br>XXXXXX | Visit * XXXXXXX | XX<br>DDMMMYYYY/ | XXXXXX | XXXXXXXX (I) | XXXXXXX | XXXXXX | XX.XXX |
| | | XXXXXXX | XX<br>DDMMMYYYY/<br>XX | XXXXXX | XXXXXXX | XXXXXXX (W) | XXXXXXX | XX.XXX |
| | | XXXXXXX | DDMMMYYYY/<br>XX | XXXXXX | XXXXXXXX (U) | XXXXXXX | XXXXXXX | XX.XXX |

Etc..

Note: \* Entry Visit is at entry to AMB114588.

I=Improved, W=Worsened, U=Unchanged

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

|-----|--------------|-----------|

Protocol: AMB114588

Population: Safety


Treatment: Ambrisentan 2.5mg

Listing 3.21: Listing of 12-Lead ECG Findings

| Centre ID/<br>Subject ID | Age(y)/<br>Sex/<br>Race | Visit | Visit Date/<br>Study Day | Result |
|---|---|---|---|---|
| XXXXXX/<br>XXXXXX | XX/<br>XXXXXX/<br>XXXXXX | Baseline ** Entry Visit * XXXXXXX | DDMMMYYYY/ XX DDMMMYYYY/ XX DDMMMYYYY/ XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | Etc | | |

Etc..

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

| F | RAP | CONFIDENTIAL | AMB114588 | l |
|---|-----|--------------|-----------|---|
|---|-----|--------------|-----------|---|

Listing 3.22: Listing of Endocrinology Assessments

Treatment: Ambrisentan 2,5mg

Population: Safety

| Centre ID/ | | | Endocrinology | | |
|---|---|---|---|---|---|
| Subject ID | Age(y)/ | | Assessment | | |
| | Sex/ | | Date/ | | Assessment |
| | Race | Visit | Study Day | Assessment Type | Result |
| XXXXXX/<br>XXXXXX | XX/<br>Male/ | Baseline | DDMMMYYYY/<br>XX | Testicular volume<br>Right/Left (units) | XXX / XXX |
| | XXXXXX | | | Male genital development Male pubic hair development | XXXXXXXXXX<br>XXXXXXXXXX<br>XXX |
| | | Entry<br>Visit * | DDMMMYYYY/<br>XX | Testicular volume<br>Right/Left (units) | XXX / XXX |
| | | | | Male genital development | XXXXXXXXXX<br>XXX |
| | | | | Male pubic hair | XXXXXXXXX |
| | | Etc | | dovezepmene | |
| XXXXXX/<br>XXXXXX | XX/<br>Female/ | XXXXXXX | DDMMMYYYY/<br>XX | Female breast development | XXXXXXXXXX<br>XXX |
| | XXXXXX | | | Female pubic hair | XXXXXXXXXX<br>XXX |
| | | Etc | | | |
| Etc | | | | | |
| XXXXX | Female/ | XXXXXXX | • | development Female breast development | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Note: \*\* Baseline is the last value recorded prior to start of study treatment from AMB112529.

\* Entry Visit is at entry to AMB114588.

Subjects are considered as belonging to the treatment group according to the highest dose received.

For some patients, pubertal development assessments were not repeated at 20 years of age if pubertal maturity had been reached in a previous visit.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588

Population: Safety

Listing 3.24: Listing of Pregnancy Results

Treatment: Ambrisentan 2,5mg

| Centre ID/<br>Subject ID | | | | | |
|---|---|---|---|---|---|
| | Age(y)/ | | Visit Date/ | | Subject became |
| | Race | Visit | Study Day | Result | pregnant? |
| XXXXXX/ | XX/ | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX | No |
| XXXXXX | XXXXXX/ | | XX | | |
| | XXXXXX | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX | |
| | | | XX | | |
| | | XXXXXXX | DDMMMYYYY/ | XXXXXXXXXXXX | |
| | | | XX | | |
| | | Etc | | | |

Etc..

Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Protocol: AMB114588


Population: Safety

Listing 3.25: Listing of Endocrinology Parameters - 20 Year Visit

Treatment: Ambrisentan 2,5mg

| Centre | Age(y)/ | 20 Year Visit | Endocrine | Assessment Type | Assessment | | |
|---|---|---|---|---|---|---|---|
| ID/ | Sex/ | Date/ | Assessment | | Result | | |
| Subject | Race | 20 Year Visit | Date/Day | | | | |
| ID | | | | | | Convert | ted Data |
| | | | | | | Value | Normal Range |
| XXXXXX/ | XX/ | DDMMMYYYY/ | DDMMMYYYY/ | Total Testosterone | XXXXXXXXXXX | | |
| XXXXXX | XXXXXX/ | 20 Years Old | XX | | | | |
| | XXXXXX | | DDMMMYYYY/ | Luteinizing Hormone | XXXXXXXXXXXX | XXX | XXX - XXX |
| | | | XX | | | | |
| | | | DDMMMYYYY/ | etc. | XXXXXXXXXXXX | XXX | XXX - XXX |
| | | | XX | | | | |
| | | | | | | XXX | XXX - XXX |
| XXXXXX/ | XX/ | DDMMMYYYY/ | DDMMMYYYY/ | Total Testosterone | XXXXXXXXXXXX | XXX | XXX - XXX |
| XXXXXX | XXXXXX/ | 20 Years Old | XX | | | | |
| | XXXXXX | | DDMMMYYYY/ | Luteinizing Hormone | XXXXXXXXXXXX | XXX | XXX - XXX |
| | | | XX | | | | |

Note: Endocrinology assessments are only displayed for subjects who completed their 20-year visit and for which endocrinology parameters are available.

USER ID: Directory/Program.sas Date Time

**Programming notes:** a listing that only include those subjects with a 20 Year Old Visit have the columns below i.e the ID/Sex/Last Visit Date/Last Visit Visit with Endo labs and the date, and then all the endo labs on that date.

Listing of and all Endo labs on that date - endocrine parameters (Follicle Stimulating Hormone, Luteinizing Hormone, Sex Hormone Binding Globulin, Total Testosterone and Inhibin B)

Population: Intent-to-Treat

Listing 3.26
Country Level Listing of Start Dates of COVID-19 Pandemic Measures

| Country | Pandemic Measures<br>Start Date |
|-------------|---------------------------------|
| Overall [1] | 2020-01-01 |
| Italy | 2020-01-01 |
| Germany | 2020-02-12 |
| etc | 2020-03-12 |

[1] The Overall row reflects the earliest pandemic measures start date. /Directory/program.sas 01JAN2002 12:01

Programming Note: Please list participating countries only

Population: Intent-to-Treat

Listing 3.27

Listing of Visits and Assessments Impacted by COVID-19 Pandemic

Site Id.: PPD
Country: Brazil

| Treatment | Unique Subject<br>Id./<br>Subject Id. | Impacted<br>Visit | Impact | Primary Reason for Impact |
|---|---|---|---|---|
| Trt A | / PPD | Visit 6 | MISSED VISIT | SUBJECT RELATED IMPACT [2] |
| | | Visit 7 | REMOTE VISIT WITH NO ASSESSMENTS MISSED | SITE RELATED IMPACT [3] |
| Trt B | | Visit 4 | SITE VISIT WITH ONE OR MORE ASSESSMENTS<br>MISSED | SITE RELATED IMPACT [3] |
| | | Visit 5 | MISSED VISIT | SUBJECT ACQUIRED COVID-19 INFECTION [1] |

<sup>[1]</sup> Subject acquired COVID-19 includes suspected, probable and confirmed.

/Directory/program.sas 01JAN2002 12:01

<sup>[2]</sup> Subject related impact include subject discretion and travel restrictions.

<sup>[3]</sup> Site related impacts include site temporarily closed, site staff unavailable, and study drug unavailable.

| RAP | | | CONFI | DENTIAL | AMB114588 | |
|---|---|---|---|---|---|---|
| Protocol: AM | IB114588 | / | | | | |
| opulation: | Safety | | | | | |
| | | | | Listing 3.28 | | |
| | List | ing of COVID-19 Ass | essments and | Symptom Assessments for Subjects | with COVID-19 Adverse Events | |
| reatment: > | | | | | | |
| Centre ID/<br>Subject ID | Adverse Event | AE Start Date | COVID-19<br>Case<br>Diagnosis<br>[1] | COVID-19 Test Performed/ Test<br>Date/<br>Results | Assessments and Symptom Assessments | Result |
| xxxxxx/<br>xxx | Coronavirus infection | 2020-04-16 | Suspected | Yes/<br>2020-04-17/<br>Indeterminate | Travel to Location with Community Transmission [2] | No |
| | | | | | Visited Health Care Facility [2] | No |
| | | | | | Contact with COVID-19 Confirmed/Probable<br>Case [2] | Unknown |
| | | | | | Medication Taken to Treat COVID-19 | Yes |
| | | | | | Fever | Yes |
| | | | | | Home Quarantined/Isolated | Unknown |
| | COVID-19 pneumonia | 2020-05-20 | Confirmed | Yes/<br>2020-05-22<br>Positive | Travel to Location with Community Transmission [2] | Yes |
| | | | | | Visited Health Care Facility [2] | No |
| | | | | | Contact with COVID-19 Confirmed/Probable<br>Case [2] | Yes |
| | | | | | Medication Taken to Treat COVID-19 | No |
| | | | | | Sore Throat | No |
| | | | | | Loss of Smell | Unknown |
| | | | | | Loss of Taste | No |
| | Coronavirus infection | 2020-04-16 | Probable | Yes/<br>2020-04-17/<br>Indeterminate | Travel to Location with Community Transmission [2] | Yes |
| | | | | | Visited Health Care Facility [2] | No |
| | | | | | Contact with COVID-19 Confirmed/Probable<br>Case [2] | Yes |
| | | | | | Medication Taken to Treat COVID-19 | No |
| | | | | | Fever | Yes |
| | | | | | Cough | Yes |
| | | | | | Asymptomatic | No |
| | | | | | Home Quarantined/Isolated | Yes |
| 1] COVID-19 C | ase Diagnosis is based on WI | HO Definition as of dd-mmr | n-yyyy | | | • |
| 2] Within 14 day | s prior to symptom onset. | | | | | |
| Directory/progra | m.sas 01JAN2002 12:01 | | | | | |

Programming Note: The COVID-19 AE terms include: Asymptomatic COVID-19, Coronavirus infection, COVID-19, COVID-19 pneumonia, Suspected COVID-19. Note that the number of COVID-19 AE terms may change


Population: Safety

Figure 3.1: Kaplan-Meier Survival Curves with 95% Confidence Bands of Time to First Treatment-Emergent Adverse Event



Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Change Treatment Labels. Also present Total group. Annotate to display number of events in each group also.

|----------------------------|
|----------------------------|

Population: Safety

Figure 3.3: Bar Chart of Treatment-Emergent Adverse Events Occurring in Two or More Subjects in any Treatment Group



Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Change Treatment Labels. Also present Total group. Continue for each preferred term.


Figure 3.4: Box plots of Haematology Data by Visit (Selected Parameters)

Parameter = <Parameter (units)>



Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Population: Safety

Programming notes: Change Treatment Labels. Also present Total group. Label vertical axes with parameter name and units. Label horizontal axis with appropriate visit structure. Repeat for each parameter. Haematology parameters (haemoglobin, hematocrit, platelets), Chemistry parameters (Total bilirubin, AST, ALT, GGT, Creatinine). Use log scale for Plasma NT-Pro BNP (Figures 2.7 and 2.8).

Protocol: AMB114588


Population: Safety

Figure 3.8: Patient Profiles of Liver Function Tests



Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Programming notes: Change Treatment Labels. Also present Total group. Present parameters ALT, AST, Alk. Phos, Total Bilirubin. Present one patient per page only, not grid of 4 patients.


Figure 3.11: Line plots of Endocrinology Assessments by Subject



Note: Subjects are considered as belonging to the treatment group according to the highest dose received.

USER ID: Directory/Program.sas Date Time

Population: Safety

Programming notes: Only one patient on a page, with a grid of plots on each page for each parameter. For Figure 3.11, plot female breast development and pubic hair development; male testicular volume, genital development and pubic hair development and change from baseline in male testicular volume (left and right separately). For Figure 2.9 (Japanese subset) plot echocardiogram parameters. For coded data, plot the numeric code and present codes on first page of the plot.

|-----|--------------|-----------|
|-----|--------------|-----------|

## 20. APPENDICES

## 20.1. Appendix 1 – IDSL Age Calculation

## IDSL standard/GSK standard of the derivation of AGE:

For this study, it was decided that the AGE is calculated based on the date of the baseline visit ie. AGEREFDT = Date of record with VISITNUM=20 in the VISIT dataset. BIRTHDT = derived by DM in DEMO dataset which contains imputed date for date of birth (ie. 30JUNYYYY).